#### The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

| Title | : | Reporting and Analysis Plan for Open-label, Dose-escalation<br>Study to Evaluate the Safety, Tolerability, Pharmacokinetics<br>and Pharmacodynamics of Single Doses of GSK2586881 in<br>Participants with Pulmonary Arterial Hypertension |
|---|---|---|
| <b>Compound Number</b> | : | GSK2586881 |
| <b>Effective Date</b> | : | 15-FEB-2018 |

#### **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 206246.
- This RAP is intended to describe the safety, pharmacodynamic and pharmacokinetic analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Interim Analyses and Statistical Analysis Complete (SAC) deliverable.

## **RAP Author(s):**

| Approver | Date | Approval<br>Method |
|---|---|---|
| PPD | | |
| Principal Statistician (Respiratory, Clinical Statistics) | | |
| Manager (Respiratory, Clinical Pharmacology) | 07-FEB-2018 | Pharma<br>TMF |

## The GlaxoSmithKline group of companies

## **RAP Team Approvals:**

| Approver | Date | Approval<br>Method |
|---|---|---|
| Director, Discovery Medicine (Respiratory TAU) | 07-FEB-2018 | Pharma TMF |
| GSK Fellow, Translational Pharmacology<br>Manager (Respiratory TAU) | 09-FEB-2018 | Pharma TMF |
| SERM Director (GCSP) | 14-FEB-2018 | Pharma TMF |
| Translational Pharmacology Manager (Respiratory TAU) | 09-FEB-2018 | Pharma TMF |
| Principal Clinical Research Scientist (CPSSO) | 07-FEB-2018 | Pharma TMF |
| Principal Data Manager (CPSSO) | 07-FEB-2018 | Pharma TMF |
| Programming Manager (Clinical Programming) | 14-FEB-2018 | Pharma TMF |

## **Clinical Statistics and Clinical Programming Line Approvals:**

| Approver | Date | Approval<br>Method |
|---|---|---|
| Director (Respiratory, Clinical Statistics) | 08-FEB-2018 | Pharma TMF |
| Director (Clinical Programming) | 15-FEB-2018 | Email |

## **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | INTRO | ODUCTION | 6 |
| 2. | SLIMA | MARY OF KEY PROTOCOL INFORMATION | 6 |
| ۷. | 2.1. | Changes to the Protocol Defined Statistical Analysis Plan | |
| | 2.1. | Study Objective(s) and Endpoint(s) | |
| | 2.3. | Study Objective(s) and Endpoint(s) | |
| | 2.4. | Statistical Hypotheses / Statistical Analyses | |
| 3. | PLAN | NED ANALYSES | 9 |
| | 3.1. | Interim Analyses | 9 |
| | 3.2. | Final Analyses | 11 |
| 4. | | YSIS POPULATIONS | |
| | 4.1. | Protocol Deviations | 11 |
| 5. | | SIDERATIONS FOR DATA ANALYSES AND DATA HANDLING<br>/ENTIONS | 19 |
| | 5.1. | Study Treatment & Sub-group Display Descriptors | |
| | 5.2. | Baseline Definitions | |
| | 5.3. | Other Considerations for Data Analyses and Data Handling Conventions | |
| | | Conventions | 10 |
| 6. | STUD | Y POPULATION ANALYSES | 14 |
| | 6.1. | Overview of Planned Study Population Analyses | 14 |
| | 6.2. | Concomitant Medications for PAH | 14 |
| 7. | PHAR | RMACODYNAMIC AND BIOMARKER ANALYSES | 15 |
| | 7.1. | Primary Analyses | 15 |
| | | 7.1.1. Endpoint / Variables | |
| | | 7.1.2. Summary Measure | |
| | | 7.1.3. Population of Interest | |
| | | 7.1.4. Strategy for Intercurrent (Post-Randomization) Events | 15 |
| | | 7.1.5. Statistical Analyses / Methods | 16 |
| | | 7.1.5.1. Statistical Methodology Specification | 16 |
| | 7.2. | Secondary Analyses | |
| | | 7.2.1. Endpoint / Variables | 18 |
| | | 7.2.2. Summary Measure | 18 |
| | | 7.2.3. Population of Interest | |
| | | 7.2.4. Strategy for Intercurrent (Post-Randomization) Events | 18 |
| | | 7.2.5. Statistical Analyses / Methods | |
| 8. | | TY ANALYSES | |
| | 8.1. | Adverse Events Analyses | |
| | 8.2. | Clinical Laboratory Analyses | |
| | 8.3. | Other Safety Analyses | 20 |
| 9. | | RMACOKINETIC ANALYSES | |
| | 9.1. | Pharmacokinetic Analyses | 21 |

| | | 9.1.1. | Endpoint / Variables | 21 |
|---|---|---|---|---|
| | | | 9.1.1.1. Drug Concentration Measures | |
| | | | 9.1.1.2. Derived Pharmacokinetic Parameters | |
| | | 9.1.2. | Population of Interest | |
| | | 9.1.3. | Statistical Analyses / Methods | 22 |
| 10. | POPU | LATION F | PHARMACOKINETIC (POPPK) ANALYSES | 23 |
| 11 | | | NETIC / PHARMACODYNAMIC ANALYSES | 24 |
| 11. | FHARI | WACOKII | NETIC / PHARIMACODTNAMIC ANALTSES | 24 |
| 12. | REFE | RENCES. | | 25 |
| 13. | APPE | NDICES | | 26 |
| | 13.1. | | x 1: Protocol Deviation Management and Definitions for | 0.0 |
| | | | e Population | |
| | 40.0 | | Exclusions from Evaluable Population | |
| | 13.2. | | x 2: Schedule of Activities | |
| | 40.0 | | Protocol Defined Schedule of Events | 27 |
| | 13.3. | | x 3: Study Phases and Treatment Emergent Adverse | 32 |
| | | 13.3.1. | Study Phases | |
| | | 13.3.1. | 13.3.1.1. Study Phases for Concomitant Medication | |
| | 13.4. | Annendi | x 4: Data Display Standards & Handling Conventions | |
| | 10.4. | 13.4.1. | Reporting Process | |
| | | 13.4.2. | Reporting Standards | |
| | | 13.4.3. | Reporting Standards for Pharmacokinetic | |
| | 13.5. | | x 5: Derived and Transformed Data | |
| | 10.0. | 13.5.1. | | |
| | | 13.5.2. | Study Population | |
| | | 13.5.3. | Pharmacodynamic and Biomarker | 36 |
| | 13.6. | | x 6: Reporting Standards for Missing Data | |
| | | 13.6.1. | Premature Withdrawals | |
| | | 13.6.2. | Handling of Missing Data | |
| | | | 13.6.2.1. Handling of Missing and Partial Dates | |
| | 13.7. | Appendix | x 7: Values of Potential Clinical Importance | |
| | | | Laboratory Values | |
| | | | ECG | |
| | | | Vital Signs | |
| | 13.8. | | x 8: Population Pharmacokinetic (PopPK) Analyses | |
| | | 13.8.1. | Population Pharmacokinetic (PopPK) Dataset | |
| | | | Specification | 42 |
| | 13.9. | Appendix | x 9: Pharmacokinetic / Pharmacodynamic Analyses | 45 |
| | | 13.9.1. | Pharmacokinetic / Pharmacodynamic Dataset | |
| | | | Specification | 45 |
| | 13.10. | | x 10: Abbreviations & Trade Marks | 64 |
| | | 13.10.1. | Abbreviations | 64 |
| | | 13.10.2. | Trademarks | 65 |
| | 13.11. | Appendix | x 11: List of Data Displays | 66 |
| | | | Data Display Numbering | |
| | | 13.11.2. | Mock Example Shell Referencing | 66 |
| | | | Deliverables | |
| | | 13.11.4. | Study Population Tables | 67 |

## 2019N405280\_00 206246

| | 13.11.5. Safety Tables | 69 |
|--------|---------------------------------------------------------|----|
| | 13.11.6. Safety Figures | |
| | 13.11.7. Pharmacokinetic Tables | |
| | 13.11.8. Pharmacokinetic Figures | 74 |
| | 13.11.9. Pharmacodynamic and Biomarker Tables | 75 |
| | 13.11.10. Pharmacodynamic and Biomarker Figures | 79 |
| | 13.11.11. Pharmacokinetic / Pharmacodynamic and Biomark | er |
| | Figures | 86 |
| | 13.11.12.ICH Listings | 89 |
| | 13.11.13. Non-ICH Listings | 91 |
| 13.12. | Appendix 13: Example Mock Shells for Data Displays | 93 |

## 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol:

| Revision Chronology: | | |
|----------------------|-------------|-------------|
| 2016N290015_00 | 04/APR/2017 | Original |
| 2016N290015_01 | 03/MAY/2017 | Amendment 1 |
| 2016N290015_02 | 07/NOV/2017 | Amendment 2 |
| 2016N290015_03 | 01/DEC/2017 | Amendment 3 |

#### 2. SUMMARY OF KEY PROTOCOL INFORMATION

## 2.1. Changes to the Protocol Defined Statistical Analysis Plan

To support internal decision making, some additional analyses have been included to output posterior probabilities for the primary hemodynamic measurements and also for Cardiac Index (CI) in relation to change from baseline (ratio to baseline).

## 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To evaluate changes in the pulmonary<br>hemodynamics after single IV doses of<br>GSK2586881 administered to<br>participants with PAH receiving<br>background PAH therapy. | Change from baseline in pulmonary vascular resistance (PVR), cardiac output (CO) and mean pulmonary artery pressure (mPAP), as data permit |
| Secondary Objectives | Secondary Endpoints |
| To evaluate the safety and tolerability of single IV doses of GSK2586881 administered to participants with PAH receiving background PAH therapy. | Adverse events (AE), clinical laboratory values, vital signs, electrocardiogram (ECG), pulse oximetry and immunogenicity. |
| To evaluate the effect of single IV doses of GSK2586881 on RAS peptide concentrations in participants with PAH receiving background PAH therapy. | Change from baseline of pulmonary wedge<br>and systemic RAS peptides<br>(e.g. Ang II, Ang(1-7), Ang(1-5) and<br>AngII/Ang(1-7) ratio) (a) |
| To evaluate the effect on biomarkers of<br>disease activity after single IV doses of<br>GSK2586881 administered to<br>participants with PAH receiving<br>background PAH therapy. | Change from baseline in NT pro-BNP, NO and cardiac troponin I. |
| To evaluate the pharmacokinetics (PK) of GSK2586881 after single IV doses of GSK2586881 in participants with PAH receiving background PAH | Plasma concentrations of GSK2586881 and derived PK parameters. |

| Objectives | Endpoints |
|---|---|
| therapy. | |
| Exploratory Objectives | Exploratory Endpoints |
| To evaluate PK/PD relationships after<br>single IV doses of GSK2586881 | RAS peptides (systemic and pulmonary wedge) and/or pulmonary vascular hemodynamic measurements compared with PK exposure. (b) |
| To evaluate pharmacogenetics (PGx). | Evaluate I/D polymorphisms in the Angiotensin<br>Converting Enzyme (ACE) gene and analyze<br>the impact on Ang II (and possibly other RAS<br>peptides), and responses to GSK2586881<br>administration. |

- (a) Note for reporting the terms 'venous (systemic) RAS peptides' and 'pulmonary wedge RAS peptides' will be presented to clearly distinguish between the systemic venous sampling and the arterial venous pulmonary wedge sampling.
- (b) Note this endpoint has been updated slightly from the current protocol amendment which states "Pulmonary wedge RAS peptides, and/or pulmonary vascular hemodynamic measurements compared with PK exposure" to clarify that both venous (systemic) and pulmonary wedge RAS data will be evaluated.

## 2.3. Study Design



## 2.4. Statistical Hypotheses / Statistical Analyses

There are no statistical hypotheses for this study. Data will be presented descriptively with supportive posterior probabilities for selected hemodynamic endpoints in relation to changes from baseline (ratio to baseline).

#### 3. PLANNED ANALYSES

## 3.1. Interim Analyses

The planned dose levels for the study are 0.1 mg/kg, 0.2 mg/kg, 0.4 mg/kg and 0.8 mg/kg. Each cohort will recruit a minimum of 4 subjects to a dose level. After the final participant has completed dosing within a given cohort and data are available, a dose escalation meeting will take place. If additional participants are added to a particular dose level, a further meeting may be held to review the additional data.

The study review team may include the following (or delegates as appropriate): Clinical Statistics, CPMS, GCSP, CIL, OSL, Medical Monitor and DQL. Other functions may be invited as required. The data will be used to support the decision to move to the next dose level as planned. Decisions made at each meeting in relation to a given dose, will be documented in the CPSR. For dose escalation decision making, the data to be reviewed will be preliminary safety, PK and hemodynamics. RAS peptide data, if available, will also be reviewed in stream.

Prior to each dose escalation meeting, unblinded safety data for this open-label study will be made available to the study team via listings from Inform and Q2 Results Viewer. In addition, CPMS will obtain the interim unblinded PK concentration data from SMS2000 via HARP according to current working practices. If any process changes occur which affect the way in which SMS2000 data is obtained during the study, then the applicable process at the time will be followed and any changes in processes between dose escalations will be documented. Descriptive tabular summaries (geometric mean, CV(%), median and range) for PK parameters and graphical presentation of PK concentration data will be produced, as appropriate, based on nominal times.

Preliminary hemodynamic data for the primary endpoints PVR, CO, mPAP and also Cardiac Index (CI) will be summarised descriptively by the Statistics and Programming team (S&P). Summary statistics and a data listing will be produced by endpoint, for each dose escalation review. In addition, a graphic will be produced for each endpoint, displaying all subjects within the given dose group, by timepoint (i.e. overlaid time profiles for each subject).

To support internal team decision making (particularly around the lower doses of 0.1 mg/kg and 0.2 mg/kg), a Bayesian analysis of change from baseline (ratio to baseline) in PVR, CO, mPAP and CI will be performed and posterior probabilities produced (see Section 7.1.5). Only analyses carried out at the final reporting effort, once all dose groups have completed, will be included in the CPSR. In addition, for the hemodynamic parameters and available RAS data, individual participant profiles may be presented alongside profiles from a previous investigator led study (NCT01884051) for visual comparison.

A summary of the dose escalation meetings is provided in the table below. The steps below assume no changes to the planned doses, however, there is flexibility to adapt/change a dose if required during the study and the format of the dose escalations below would be modified to accommodate any dose changes. In addition, flexibility is

allowed within the study to recruit additional participants to a previous cohort (post dose escalation review) if a need for further data is required. Any additional participants would be summarised as part of the final (all dose groups) reporting.

| Dose Escalation [DE] Level | Data to be Reviewed/Output after a minimum of 4 participants have completed |
|---|---|
| Review of Dose Level 1: 0.1 mg/kg (planned) DE[1] | <ul> <li>Safety: Via Q2 Results Viewer and Inform</li> <li>PK: CPMS to use SMS2000 data based on nominal times and generate summaries, and graphs.</li> <li>PD (PVR, CO, mPAP &amp; CI): S&amp;P will generate a summary table, listing and individual subject graphic (all subjects on one graph) for each endpoint based on SI data provided by Data Management via HARP. Outputs may be produced using PC SAS or HARP.</li> <li>Posterior probabilities (PVR, CO, mPAP &amp; CI).</li> <li>Review of RAS data (if available or post dose escalation meeting).</li> </ul> |
| <ul> <li>Review of Dose Level 2: 0.2 mg/kg (planned)</li> <li>DE[2]</li> </ul> | <ul> <li>Safety: Via Q2 Results Viewer and Inform</li> <li>PK: CPMS to use SMS2000 data based on nominal times and generate summaries, and graphs.</li> <li>PD (PVR, CO, mPAP &amp; CI): S&amp;P will generate a summary table, listing and individual subject graphic (all subjects on one graph) for each endpoint based on SI data provided by Data Management via HARP. Outputs may be produced using PC SAS or HARP.</li> <li>Posterior probabilities (PVR, CO, mPAP &amp; CI).</li> <li>Review of RAS data (if available or post dose escalation meeting)</li> </ul> |
| <ul> <li>Review of Dose Level 3: 0.4 mg/kg (planned)</li> <li>DE[3]</li> </ul> | <ul> <li>Safety: Via Q2 Results Viewer and Inform</li> <li>PK: CPMS to use SMS2000 data based on nominal times and generate summaries, and graphs.</li> <li>PD (PVR, CO, mPAP &amp; CI): S&amp;P will generate a summary table, listing and individual subject graphic (all subjects on one graph) for each endpoint based on SI data provided by Data Management via HARP. Outputs may be produced using PC SAS or HARP.</li> <li>Posterior probabilities (PVR, CO, mPAP &amp; CI).</li> <li>Review of RAS data (if available or post dose escalation meeting)</li> </ul> |
| Final Reporting (SAC) | Data for all dose levels including the planned 4 <sup>th</sup> dose of 0.8 mg/kg will be summarised in the final reporting. |

## 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All participants have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release (DBR) and database freeze (DBF) has been declared by Data Management.
- 3. All criteria for unblinding the randomization codes have been met (*the study is openlabel but randomisation numbers are still generated for each cohort*).
- 4. Randomization codes have been distributed according to RandAll NG procedures (the study is open-label but a Randall dataset is still generated)

#### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses<br>Evaluated |
|---|---|---|
| Enrolled | All participants who sign the ICF | Screening summaries |
| Safety | All participants who take at least 1 dose of study treatment. Participants will be analysed according to the treatment they actually received. | Study Population & Safety |
| Evaluable | Evaluable: All participants who are in the Safety population who complete all Day 1 assessments (including up to 24 hours post dose) and were not deemed to have had major protocol deviations (as defined within the PDMP) | PD |
| Pharmac-<br>okinetic | Subjects in the 'Safety' population for whom a pharmacokinetic sample was obtained and analysed. | PK |

Refer to Appendix 11: List of Data Displays which details the population used for each display.

#### 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.

- Data will be reviewed prior to freezing the database to ensure all important deviations and deviations which may lead to exclusion from the analysis are captured and categorised on the protocol deviations dataset.
- o This dataset will be the basis for the summaries and listings of protocol deviations.
- A separate listing of all inclusion/exclusion criteria deviations will also be provided.
   This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

## 5.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions | | | |
|---|---|---|---|
| Rar | ndAll NG | Data Displays for | Reporting |
| Code | Description | Description | Order in TLF |
| Α | Dose 1 | GSK2586881 i.v. 0.1 mg/kg | 1 |
| В | Dose 2 | GSK2586881 i.v. 0.2 mg/kg | 2 |
| С | Dose 3 | GSK2586881 i.v. 0.4 mg/kg | 3 |
| D | Dose 4 | GSK2586881 i.v. 0.8 mg/kg | 4 |

**NOTES:** Order represents treatments being presented in TFL, as appropriate.

As this is a small study, for graphical representation, each participant may be assigned a unique combination of plotting symbol / line style / colour based on the attribute map facility using SAS SG procedures. The GSK statistician will provide further details to the study team. The unique characterisation will apply to all graphics of by subject data. In the case that an alternative statistical package is used, every effort will be made to apply a unique set of graphical characterisations for subjects.

In addition, for graphics summarising data by dose group, colours/symbols for each dose group will be made consistent throughout. For example:

GSK2586881 i.v. 0.1 mg/kg - blue diamond GSK2586881 i.v. 0.2 mg/kg - red square GSK2586881 i.v. 0.4 mg/kg - green circle GSK2586881 i.v. 0.8 mg/kg - black star.

#### 5.2. Baseline Definitions

For all endpoints (except as noted in baseline definitions) the baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. If time is not collected, Day 1 assessments are assumed to be taken prior to first dose and used as baseline.

| Parameter | _ | nents Considered As<br>aseline | Baseline Used in Data<br>Display |
|---|---|---|---|
| | Screening | Day 1 (Pre-Dose) | |
| Safety | | | |
| Labs | Х | X | Day 1 |
| ECGs | X [1] | X [1] | Day 1 [1] |
| Vital Signs | X [1] | X | Day 1 |
| Pulse Oximetry | Х | X | Day 1 |
| Immunogenicity | | Х | Day 1 |

| Parameter | • | nents Considered As<br>aseline | Baseline Used in Data<br>Display |
|---|---|---|---|
| | Screening | Day 1 (Pre-Dose) | |
| Biomarkers/Pharmacodynamic | | | |
| RAS peptides, disease activity biomarkers | | X | Day 1 |
| Hemodynamics (e.g., PVR, CO, mPAP & CI) | | Х | Day 1 |

<sup>[1]</sup> Unless otherwise stated, the mean of replicate assessments at any given time point will be used as the value for that time point.

Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing.

## 5.3. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---------|----------------------------------------------------------------|
| 13.3 | Appendix 3: Study Phases and Treatment Emergent Adverse Events |
| 13.4 | Appendix 4: Data Display Standards & Handling Conventions |
| 13.5 | Appendix 5: Derived and Transformed Data |
| 13.6 | Appendix 6: Reporting Standards for Missing Data |
| 13.7 | Appendix 7: Values of Potential Clinical Importance |

#### 6. STUDY POPULATION ANALYSES

## 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the Safety population, unless otherwise specified.

Study population analyses including analyses of subject's disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, and exposure and treatment compliance will be based on GSK Core Data Standards. Data collected for functional class, 6-minute walking distance and PAH underlying cause will also be summarised. Details of the planned displays are presented in Appendix 11: List of Data Displays.

#### 6.2. Concomitant Medications for PAH

PAH medications (reason for medication) will be reviewed by the medical monitor. Two reviews will be planned; one prior to DBF to enable pre-programming and a final review on receipt of final concomitant medication data at DBF. An intermediate review will take place if required. A spreadsheet of the databased concomitant medications will be generated by S&P for review by the medical monitor, who will add a flag to records that are relevant to PAH. S&P will then use the spreadsheet when creating the derived A&R CMANAL dataset to include the flagged records for use within the corresponding output.

In addition, to support the programming of PCI ranges for International Normalized Ratio (INR), Prothrombin time (PT) and PTT (see Section 13.7.1) medications of Heparin or Warfarin will need to be confirmed per participant by review of related concomitant medication terms. This will require non-standard coding for the programming of PCI ranges.

### 7. PHARMACODYNAMIC AND BIOMARKER ANALYSES

## 7.1. Primary Analyses

#### 7.1.1. Endpoint / Variables

The primary endpoints are hemodynamic measurements of:

- Pulmonary Vascular Resistance (PVR)
- Cardiac Output (CO)
- Mean Pulmonary Artery Pressure (mPAP)

Additional hemodynamic endpoints are:

- Right Atrial Pressure
- Pulmonary Artery Systolic Pressure
- Pulmonary Artery Diastolic Pressure
- Pulmonary Capillary Wedge Pressure
- Cardiac Index (CI)
- Pulmonary Artery Oxygen Saturation

## 7.1.2. Summary Measure

Absolute and change from baseline will be the summary measures of interest for hemodynamic endpoints. Hemodynamic measurements will also be log transformed to aid further analysis and therefore the change from baseline geometric means at each post-dose timepoint, will represent a percentage increase/decrease from baseline (presented as a ratio to baseline).

#### 7.1.3. Population of Interest

The primary efficacy analyses will be based on the Evaluable population, unless otherwise specified.

#### 7.1.4. Strategy for Intercurrent (Post-Randomization) Events

Hemodynamic data will be collected according to the timepoints referenced in Appendix 2: Schedule of Activities. Missing data will not be replaced.

The Evaluable population defined in Section 4, utilises patients who complete all Day 1 assessments. If a consistent pattern of withdrawals prior to the completion of Day 1 is noted (for example, sensitivity to the catheter causing it to be removed early) which causes a lower than expected Evaluable population, then additional reviews of available data for those not included in the Evaluable population may take place.

### 7.1.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 11: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

A Bayesian analysis will be conducted by dose group and timepoint displaying posterior probabilities as detailed in Section 7.1.5.1.

#### 7.1.5.1. Statistical Methodology Specification

#### **Endpoint / Variables**

PVR, CO, mPAP and CI

#### **Model Specification**

- The description below describes the current thinking of how to analyse this endpoint. The
  proposed model will be assessed, and if not appropriate alternative models could be used.
  Reasons for and a full description of alternative modeling/analysis methods used would be fully
  documented in the CPSR.
- Separate Bayesian repeated measures mixed effect models (one model per endpoint) will be
  used to assess changes from baseline for dose group and post-treatment timepoint
  combinations. Individual patient data will be log-transformed prior to analysis and change from
  baseline (CFB) calculated on transformed data. The Baseline values (BS) used in the model
  should also have been log-transformed prior to their use.

Note: The modeling described below should be appropriately modified for the 1<sup>st</sup> interim analysis (e.g. to remove terms involving dose).

Response: CFB = BS\*Time + Time + Dose + Dose\*Time

Fixed effects: (class) Time [3 levels, 1H, 2H and 4H], Dose level [either 0.1, 0.2, 0.4 or 0.8

mg/kg as appropriate to the timing of the <interim> analysis].

Fixed effects: (continuous): Baseline value (on the Ln scale)

Repeated measures on Time, Subject=Subject, Unstructured Variance Co-Variance (VCV)

matrix (3x3)

Appropriate combinations of the fitted model parameters will be used to obtain posterior distributions (one per planned comparison). The planned comparisons are the equivalent of the LSMeans for each timepoint within each dose level (on a back transformed scale their interpretation is the fold change c.f. baseline).

- Non-informative priors should be assumed for all model parameters. Therefore, unless there is
  a large proportion of missing data, the posterior probabilities may be obtained by fitting the
  proposed model using SAS PROC MIXED and extracting the appropriate pieces of
  information.
- However, if PROC MCMC is used then the default prior for each fixed effect model parameter should be Normal~(Mean=0, Var=1E6). The default prior for the VCV matrix would be an Inverse-Wishart with parameters k and S (where S = (k p 1) \* R and p = dimension of the

VCV matrix). Under this framework  $\bf R$  can be thought of as a best guess for the VCV of the endpoint being modelled. Care should be taken in the choice of  $\bf k$  and  $\bf R$  for each endpoint. The default should set  $\bf k$  = 5 (p + 2) and  $\bf R$  should be set to the following for each endpoint, in order to obtain the value of  $\bf S$  to put into the inverse-Wishart prior:

| CO (L/min) | CI (L/Min/m**2) | PVR (Wood units) | mPAP (mmHg) |
|---|---|---|---|
| $ \begin{pmatrix} 0.160 & 0.096 & 0.017 \\ 0.096 & 0.064 & 0.014 \\ 0.017 & 0.014 & 0.005 \end{pmatrix} $ | 0.160 0.096 0.017 0.096 0.064 0.014 0.017 0.014 0.005 | (0.323 0.204 0.070 0.204 0.544 0.111 0.070 0.111 0.030 | $ \begin{pmatrix} 0.031 & 0.031 & 0.007 \\ 0.031 & 0.039 & 0.017 \\ 0.007 & 0.017 & 0.018 \end{pmatrix} $ |

These values of **R** were obtained from a historical study (GSK ID 204696) and unit conversion may be required to match this study.

(Note: depending on the software used and parameterization the above may need to be adjusted to use a Wishart instead of the inverse-Wishart).

Given the small sample sizes in this study the above priors may be more informative/influential than intended. An optional sanity check may be made by comparing the observed sample VCV matrix to the prior. If there are large discrepancies alternative priors may be attempted/evaluated as part of sensitivity analyses (and the output from the most appropriate model reported in the CPSR along with a brief justification/discussion on any switched priors). For example **R** may be replaced by the observed sample VCV matrix (on the log transformed scale) once the study data are available.

- Posterior medians and 95% credible intervals will be presented for each posterior distribution.
   As stated previously estimates will be back-transformed so that the difference from baseline represents a ratio.>
- The posterior distributions will be used to produce several probability statements, presented in tabular format. This will include but are not limited to:
  - PVR, the probability of any % reduction from baseline (<0%), <-20% and <-30% (equivalent to <1, <0.8 and <0.7 in terms of a ratio from baseline)
  - CI, the probability of any % increase from baseline (>0%), >20% and >30% (equivalent to >1, >1.2 and >1.3 in terms of a ratio from baseline)
  - CO probability of >0% increase (or >1 in terms of a ratio from baseline)
  - mPAP probability of <0% (or <1 in terms of a ratio from baseline)

#### **Model Checking & Diagnostics**

Assumptions regarding normality will apply if the analysis is conducted using proc mixed.
 Should major violations occur (caveat being that the sample sizes will be small) then a non-parametric Wilcoxon signed rank test may be considered.

#### **Model Results Presentation**

A summary table will be produced for each endpoint by dose group and timepoint, displaying
medians and 95% credible intervals for the change from baseline (ratio to baseline) endpoints
along with the posterior probabilities as described above.

## 7.2. Secondary Analyses

#### 7.2.1. Endpoint / Variables

The secondary biomarker endpoints are:

Venous (systemic) RAS Peptides:

- Ang II
- Ang(1-7)
- Ang(1-5)
- Ang II / Ang(1-7)

Pulmonary Wedge RAS Peptides:

- Ang II
- Ang(1-7)
- Ang(1-5)
- Ang II / Ang(1-7)

Disease Activity Biomarkers:

- NT pro-BNP
- Serum NO
- Cardiac troponin I

#### 7.2.2. Summary Measure

Absolute and change from baseline will be the summary measures of interest for RAS Peptides and Disease Activity Biomarkers. As a log-transformed summary for biomarkers will be included, the change from baseline geometric means will represent a percentage increase/decrease from baseline (presented as a ratio to baseline).

#### 7.2.3. Population of Interest

The secondary analyses will be based on the Evaluable population, unless otherwise specified.

#### 7.2.4. Strategy for Intercurrent (Post-Randomization) Events

Venous (systemic) RAS peptide data will be collected at timepoints in line with the PK. Pulmonary wedge RAS peptides will be collected in line with hemodynamic data predose to 4 hours post dose. Disease activity biomarkers will be collected at timepoints up to 24 hours. For details on data collection timepoints, refer to Appendix 2: Schedule of Activities. Missing data will not be replaced but data recorded as NQ will be imputed based on details given in Appendix 6: Reporting Standards for Missing Data.

## 7.2.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 11: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.2.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

## 8. SAFETY ANALYSES

The safety analyses will be based on the Safety population, unless otherwise specified.

## 8.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs), Serious (SAEs) and other significant AEs will be based on GSK Core Data Standards. The details of the planned displays are provided in Appendix 11: List of Data Displays.

## 8.2. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Hematology laboratory tests, Urinalysis, and liver function tests will be based on GSK Core Data Standards. The details of the planned displays are in Appendix 11: List of Data Displays.

## 8.3. Other Safety Analyses

The analyses of non-laboratory safety test results including ECGs and vital signs will be based on GSK Core Data Standards, unless otherwise specified. The details of the planned displays are presented in Appendix 11: List of Data Displays.

For systolic blood pressure (SBP), diastolic blood pressure (DBP) and heart rate (HR), in addition to standard tables and listings, the change from baseline over time by dose group will displayed graphically along with individual subject profiles.

#### 9. PHARMACOKINETIC ANALYSES

## 9.1. Pharmacokinetic Analyses

### 9.1.1. Endpoint / Variables

#### 9.1.1.1. Drug Concentration Measures

Refer to Appendix 4: Data Display Standards & Handling Conventions (Section 13.4.3 Reporting Standards for Pharmacokinetic).

#### 9.1.1.2. Derived Pharmacokinetic Parameters

Pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin Pro. For the final reporting effort (see Section 3.1 for interim details of pharmacokinetic analyses), all calculations of non-compartmental parameters will be based on actual sampling times. Pharmacokinetic parameters listed will be determined from the plasma concentration-time data, as data permits.

| Parameter | Parameter Description |
|---|---|
| AUC(0-t) | Area under the concentration-time curve from time zero to the time of the last quantifiable concentration (C(t)) will be calculated using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid. |
| AUC(0-∞) | Area under the concentration-time curve extrapolated to infinity will be calculated as: AUC = AUC(0-t) + C(t) / lambda_z |
| Cmax | Maximum observed concentration, determined directly from the concentration-time data. |
| tmax | Time to reach Cmax, determined directly from the concentration-time data. |
| t½ | Apparent terminal half-life will be calculated as: t½ = ln2 / lambda_z |
| Clast | Last observed quantifiable concentration |
| tlast | Time of the last observed quantifiable concentration |
| CL | Plasma clearance |
| V | Volume of distribution |
| Lambda_z | The first order rate constant associated with the terminal (log-linear) portion of the concentration-time curve. |
| Lambda_z_lower | First time point used in computing Lambda_z. |
| Lambda_z_upper | Last time point used in computing Lambda_z. |
| #pts | Number of points used in computing Lambda_z. |
| r-squared | R-squared of Lambda_z computation. |

- Additional parameters may be included as required
- Lambda\_z is the terminal phase rate constant

## 9.1.2. Population of Interest

The primary pharmacokinetic analyses will be based on the Pharmacokinetic population, unless otherwise specified.

## 9.1.3. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 11: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 9.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

# 10. POPULATION PHARMACOKINETIC (POPPK) ANALYSES

A population PK analysis, to characterize the population pharmacokinetics of GSK2586881 administered IV in participants with PAH, may be conducted, if appropriate. To support this analysis, a NONMEM-specific data file will be generated, the specifications of which are provided in Appendix 8: Population Pharmacokinetic (PopPK) Analyses. Specific details of the analysis, which may be part of a population PK meta-analysis with historical data, will be appropriately documented in a separate RAP and report which will be written by, or under the direct auspices of, Clinical Pharmacology Modelling and Simulation (CPMS), GlaxoSmithKline, as required. The timeline for these analyses will be independent of the analysis described in this RAP.

# 11. PHARMACOKINETIC / PHARMACODYNAMIC ANALYSES

The primary goal of these exploratory analyses are to investigate the pharmacokinetic / pharmacodynamic relationship(s) of GSK2586881 administered IV in participants with PAH. Graphics of RAS Peptides vs PK concentrations and hemodynamic endpoints vs PK concentrations using the PK population, unless otherwise specified, will be initially used to assess any potential relationships. If data permit, the potential association between systemic exposure of GSK2586881 and RAS peptides (Ang II, Ang(1-7), Ang(1-5) and AngII/Ang(1-7) from both venous (systemic) and pulmonary wedge sampling) and clinical endpoints (e.g., PVR, CO, mPAP and CI) may be studied. To support any analyses that is required based on the initial graphical assessment, NONMEM-specific data files will be generated, the specifications of which are provided in Appendix 9: Pharmacokinetic / Pharmacodynamic Analyses. Specific details of any PK/PD analysis, which may be part of a population PK meta-analysis with historical data. will be appropriately documented in a separate RAP and report which will be written by, or under the direct auspices of, Clinical Pharmacology Modelling and Simulation (CPMS), GlaxoSmithKline, as required. The timeline for these analyses will be independent of the analysis described in this RAP.

## 12. REFERENCES

Not Applicable

## 13. APPENDICES

# 13.1. Appendix 1: Protocol Deviation Management and Definitions for Evaluable Population

## 13.1.1. Exclusions from Evaluable Population

Subjects with major/important protocol deviations will be excluded from Evaluable Population. The Protocol Deviation Management Plan (PDMP) will be used to determine major/important protocol deviations that will lead to exclusion from the Evaluable Population.

## 13.2. Appendix 2: Schedule of Activities

## 13.2.1. Protocol Defined Schedule of Events

| Procedure | Screening<br>(up to 28<br>days | | | | Trea | tment Pe | eriod | | | | Follow-<br>up<br>Day 7-<br>14 | Follow-<br>up Day<br>28 ± 3<br>days | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | before<br>dosing) | Pre-<br>dose <sup>1</sup> | 0h | 0.08h<br>(5<br>min) <sup>2</sup> | 0.5h | 1h | 2h | 4h | 8h | 24h | | - | |
| Informed consent | X | | | | | | | | | | | | |
| Genetics consent | Х | | | | | | | | | | | | |
| Inclusion and exclusion criteria | Х | | | | | | | | | | | | Recheck clinical<br>status before<br>randomization<br>and/or 1st dose of<br>study medication |
| Demography | Х | | | | | | | | | | | | |
| Full physical examination including height and weight | Х | | | | | | | | | | | | |
| Medical history (includes<br>substance usage and<br>family history of<br>premature CV disease) | Х | | | | | | | | | | | | Substances: drugs,<br>alcohol, tobacco<br>and caffeine |
| Past and current medical conditions | Х | | | | | | | | | | | | |

| Procedure | Screening<br>(up to 28<br>days | | | | Trea | itment Pe | Follow-<br>up<br>Day 7-<br>14 | Follow-<br>up Day<br>28 ± 3<br>days | Notes | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | before<br>dosing) | Pre-<br>dose <sup>1</sup> | 0h | 0.08h<br>(5<br>min) <sup>2</sup> | 0.5h | 1h | 2h | 4h | 8h | 24h | | |
| Serum OR urine pregnancy test (WOCBP only) | X | Х | | | | | | | | | X | |
| FSH and estradiol test<br>(postmenopausal<br>females only as needed) | Х | | | | | | | | | | | |
| Human<br>Immunodeficiency Virus<br>(HIV), Hepatitis B and C<br>screening | х | | | | | | | | | | | If test performed<br>within 3 months<br>prior to first dose of<br>study treatment,<br>testing at screening<br>is not required |
| Functional classification | X | | | | | | | | | | | |
| 6 Minute Walk Distance | X3 | | | | | | | | | | | |
| Admission | | Х | | | | | | | | | | Participants may be admitted the day before dosing to enable completion of required pre-dose time point assessments. |
| Brief physical | | Х | | | | | | | | | Х | |
| Study Treatment | | | Х | | | | | | | | | |

| Procedure | Screening<br>(up to 28<br>days | | | | Trea | itment Pe | riod | | | | Follow-<br>up<br>Day 7-<br>14 | Follow-<br>up Day<br>28 ± 3<br>days | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | before<br>dosing) | Pre-<br>dose <sup>1</sup> | 0h | 0.08h<br>(5<br>min)² | 0.5h | 1h | 2h | 4h | 8h | 24h | | , | |
| Vital Signs | fital Signs X X X X X | X | X X | | x x | X | | Vital signs will be measured after 5 minutes supine at all time points. | | | | | |
| Vital Olgilo | Α | Α | | | Α | ^ | ^ | χ | ^ | ^ | X | | Triplicate blood<br>pressure (BP) will<br>be taken at<br>screening only. |
| Pulse Oximetry (SpO <sub>2</sub> ) | X | X | | | X | X | Х | X | Х | х | Х | | Pulse oximetry will<br>be measured and<br>recorded with each<br>blood pressure<br>assessment |
| Laboratory assessments<br>(include liver chemistries,<br>haematology panel and<br>coagulation panel) | X | Х | | | | | | | | х | Х | | |
| Urinalysis | Х | | | | | | | | | Х | | | |
| 12-lead ECG | Х | Х | | | | | | Х | | Х | Х | | Triplicate will be performed at Screening and Predose |

| Procedure | Screening<br>(up to 28<br>days | | | | Trea | atment Pe | riod | | | | Follow-<br>up<br>Day 7-<br>14 | Follow-<br>up Day<br>28 ± 3<br>days | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | before<br>dosing) | Pre-<br>dose <sup>1</sup> | 0h | 0.08h<br>(5<br>min) <sup>2</sup> | 0.5h | 1h | 2h | 4h | 8h | 24h | | | |
| Telemetry | | | ← | | | | | | <del>-</del> | , | | | Monitoring to start<br>30min prior to<br>treatment<br>administration and<br>continue throughout<br>the study until 24h<br>after dosing |
| Right heart catheter Insertion | | ← | | | | | | <del>-</del> | | | | | RHC inserted prior<br>to dose and<br>removed after the<br>4h hemodynamic<br>measurement |
| Blood sample for biomarkers of disease activity | | Х | | | | | х | Х | | Х | | | |
| Blood sample for Nitric<br>Oxide | | Х | | | | | Х | Х | | Х | | | |
| Blood sample for PK | | Х | | Х | Х | Х | Х | Х | Х | Х | | | |
| Blood sample for immunogenicity | | Х | | | | | | | | | Х | X | |

| Procedure | Screening<br>(up to 28<br>days | | | | Trea | Follow-<br>up<br>Day 7-<br>14 | Follow-<br>up Day<br>28 ± 3<br>days | Notes | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | before<br>dosing) | Pre-<br>dose <sup>1</sup> | 0h | 0.08h<br>(5<br>min) <sup>2</sup> | 0.5h | 1h | 2h | 4h | 8h | 24h | | |
| Blood sample for renin-<br>angiotensin system<br>biomarkers | | Х | | х | Х | Х | х | х | X | Х | Х | |
| Blood sample for transpulmonary RAS biomarkers | | Х | | | | Х | Х | Х | | | | |
| Hemodynamic measurements | | Х | | | | Х | Х | х | | | | |
| Genetic sample | | Х | | | | | | | | | | Can be taken any time after consent |
| Discharge | | | | | | | | | | Х | | |
| AE review | | ←=== | ====== | | ====== | | | | | <del>-</del> | Х | |
| SAE review | Х | <b>←===</b> | | ====== | ====== | ====> | Х | | | | | |
| Concomitant medication review <sup>4</sup> | Х | Х | | | | | | | | | Х | |

- Pre-dose measurements may be taken any time after admission up until dosing.
   Procedures will be completed immediately after dosing has completed.
- 3. If the six minute walk(6MW) has been performed in the last 6 months, and participant has been stable on current medications then there is no need to repeat. Historical data will be databased.
- 4. Concomitant medications for the 30 days prior (8 weeks prior for PAH medications) will be reviewed/recorded at screening to evaluate eligibility and changes will be recorded throughout the study.

## 13.3. Appendix 3: Study Phases and Treatment Emergent Adverse Events

## 13.3.1. Study Phases

This is a single dose study. Assessments and events will be classified according to time of occurrence relative to the start date and time of the study treatment.

| Treatment State | Definition |
|---|---|
| Pre-Treatment | AE Start Date / Time < Study Treatment Start Date / Time This will apply to all subjects enrolled into the study, including those who were not assigned to a dose (screen failures). For screening failures, any SAEs will be captured in the relevant listing. For dosed subjects included in the Safety population, these events will be captured in summary listings with treatment group='Pre-Treatment'. |
| On-Treatment | Study Treatment Start Date / Time ≤ AE Start Date / Time ≤ Follow-up (Day 7-14) Date |
| Post-Treatment | AE Start Date > Follow-Up (Day 7-14) Date There shouldn't be any instances of this. Subjects return for a follow-up visit between Days 7 and 14 and AEs/SAEs prior to this will be recorded. Subjects then return for a Day 28 follow-up but AEs/SAEs will not be recorded. |
| Onset Time Since<br>1st Dose<br>(Days/Hours/Mins) | If Study Treatment Start Date / Time ≤ AE Start Date / Time = AE Start Date / Time – Study Treatment Start Date / Time + 1 (min) Missing otherwise. A calculation to assess the time since the single dose up until the start time of the AE. Example: If Dose was administered at 08:00am 01OCT2017 and AE started at 09:10am 01OCT2017, then onset time since <b>first</b> dose would be 0d 1h 11m. |
| Duration<br>(Days/Hours/Mins) | AE Resolution Date /Time – AE Onset Date / Time + 1 (min) Example: AE started at 08:00am and resolved at 08:30am on the same day, then duration would be 0d 0h 31m |
| Drug-related | If relationship is marked 'YES' on Inform OR value is missing. |

#### 13.3.1.1. Study Phases for Concomitant Medication

| Study Phase | Definition |
|---|---|
| Prior | If medication end date is not missing and is before 28 days prior to screening visit |
| Concomitant | Any medication that is not a prior |

#### NOTES:

 Please refer to Appendix 6: Reporting Standards for Missing Data for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing.

## 13.4. Appendix 4: Data Display Standards & Handling Conventions

### 13.4.1. Reporting Process

| Software | |
|---|---|
| The currently supported versions of SAS software will be used. | |
| Reporting Area | |
| HARP Server | : \\UK1SALX00175.corpnet2.com\ARENV\ |
| HARP Compound | : \ARPROD\GSK2586881\206246\Internal_01 |
| | : \ARPROD\GSK2586881\206246\Internal_02 |
| | : \ARPROD\GSK2586881\206246\Internal_03 |
| | : \ARPROD\GSK2586881\206246\Internal_04 |
| | : \ARPROD\GSK2586881\206246\Final_01 |
| Analysis Datasets | |
| Analysis datasets will be created according to Legacy GSK A&R dataset standards. | |
| Generation of RTF Files | |
| RTF files will be generated for the final reporting effort. | |

#### 13.4.2. Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location: https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics
- Subject level listings in the main body of the GSK Clinical Study Report. All subject level listings should be located in the modular appendices as ICH or non-ICH listings

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days
    on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.

| Unscheduled Visits | |
|---|---|
| Unscheduled visits will not be included in summary tables and figures. | |
| All unscheduled visits will be included in listings. | |
| Descriptive Summary Statistics | |
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

## 13.4.3. Reporting Standards for Pharmacokinetic

| Pharmacokinetic Concentration Data | |
|---|---|
| PC Windows Non-<br>Linear (WNL) File | PC WNL file (CSV format) for the non-compartmental analysis by Clinical Pharmacology Modelling and Simulation function will be created according to GUI_51487. Note: Concentration values will be imputed as per GUI_51487 |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. Refer to IDSL Statistical Principle 6.06.1. Note: For standard PK outputs concentration values will be imputed as per GUI_51487 for descriptive summary statistics/analysis and summarized graphical displays only. For PK/PD graphics only which are generated by S&P, ½ LLQ can be used for NQ PK data to coincide with methods used for Biomarker data (see Section 13.6.2). Variables relating to different imputation methods for PK data will be available within the derived A&R PKCNC dataset. |
| NONMEM/Pop PK<br>File | Pop-PK file (CSV format) for the POP-PK analysis by Clinical Pharmacology Modelling and Simulation function will be created according to the data specification detailed in Section 13.8.1 Population Pharmacokinetic (PopPK) Dataset Specification. |
| NONMEM/PK/PD<br>File | PK/PD file (CSV format) for the PK/PD analysis by Clinical Pharmacology Modelling and Simulation function will be created according to the data specification detailed in Section 13.9.1 Pharmacokinetic/Pharmacodynamic Dataset Specification. |
| Pharmacokinetic Parameter Data | |
| Is NQ impacted PK<br>Parameters Rule<br>Being Followed | Yes, refer to [Standards for Handling NQ Impacted PK Parameters]. |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. The following PK parameters will not included in summary tables: Lambda_z, lambda_z_lower, lambda_z_upper, #pts, R squared |

### 13.5. Appendix 5: Derived and Transformed Data

#### 13.5.1. General

#### **Multiple Measurements at One Analysis Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values within a time window the value closest to the target day for that window will be used. If values are the same distance from the target, then the mean will be taken.
- Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### **Study Day**

- Calculated as the number of days from First Dose Date:
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < First Dose Date → Study Day = Ref Date First Dose Date</li>
  - Ref Data ≥ First Dose Date → Study Day = Ref Date (First Dose Date) + 1

### 13.5.2. Study Population

#### **Extent of Exposure**

- Number of days of exposure to study drug will be calculated based on the formula:
   Duration of Exposure in Days = Treatment Stop Date (Treatment Start Date) + 1
- Participants who were randomized but did not report a treatment start date will be categorised as having zero days of exposure.

### 13.5.3. Pharmacodynamic and Biomarker

#### **Pharmacodynamic**

#### **Pulmonary Hemodynamics**

Pulmonary Vascular Resistance (PVR)

[All endpoints will be provided in SI datasets]

Cardiac Output (CO)

Mean Pulmonary Artery Pressure (mPAP)

Cardiac Index (CI)
Right Atrial Pressure

Pulmonary Artery Systolic Pressure

Pulmonary Artery Diastolic Pressure

Pulmonary Capillary Wedge Pressure

Pulmonary Artery Oxygen Saturation

Variance stabilising transformations (e.g. taking natural logarithms of the observed responses) may be implemented on a per endpoint basis, if deemed necessary by the study statistician. If transformations are used the results will be reported on the back-transformed response scales. When assessing change from baseline, the individual timepoint values will be log-transformed prior to calculating a change from baseline difference (in log transformed values). Back transformation and summaries of the geometric mean and 95% CI of the back-transformed change from baseline calculations will represent percentage increase/decrease from baseline (presented as a ratio to baseline).

#### Biomarker

#### **RAS Peptides**

#### RAS Venous (systemic) Samples:

- Ang II, Ang(1-5), Ang(1-7) will be provided in SI datasets
- Ang II / Ang(1-7) ratio will be derived in A&R datasets

#### RAS Pulmonary Wedge Samples:

- Ang II, Ang(1-5), Ang(1-7) will be provided in SI datasets
- Ang II / Ang(1-7) ratio will be derived in A&R datasets

#### **Disease Activity Biomarkers**

#### NT Pro-BNP, NO and Cardiac Troponin I will be provided in SI datasets

For biomarkers, variance stabilising transformations (e.g. taking natural logarithms of the observed responses) may be implemented on a per endpoint basis, if deemed necessary by the study statistician. If transformations are used the results will be reported on the back-transformed response scales.

When assessing change from baseline, the individual timepoint values will be log-transformed prior to calculating a change from baseline difference (in log transformed values). Back transformation and summaries of the geometric mean and 95% CI of the back-transformed change from baseline calculations will represent percentage increase/decrease from baseline.
| Pharmacodyr | Pharmacodynamic | | | | | |
|---|---|---|---|---|---|---|
| Source of Bio | Source of Biomarker Data | | | | | |
| Biomarker<br>Category | Analyte | Sample | Method | Lab | Matrix | Total samples expected per subject |
| RAS | Ang II | Venous | LC/MS | Q2 | Plasma | 9 |
| Peptides <sup>1</sup> | Ang (1-5) | Venous | LC/MS | Q2 | Plasma | 9 |
| | Ang (1-7) | Venous | LC/MS | Q2 | Plasma | 9 |
| RAS<br>Peptides <sup>2</sup> | Ang II | Pulmonary<br>Wedge | LC/MS | Q2 | Plasma | 4 |
| | Ang (1-5) | Pulmonary<br>Wedge | LC/MS | Q2 | Plasma | 4 |
| | Ang (1-7) | Pulmonary<br>Wedge | LC/MS | Q2 | Plasma | 4 |
| Disease<br>Biomarkers <sup>3</sup> | NT pro-BNP | Venous | Elisa | Q2 | Serum | 4 |
| | Nitric Oxide | Venous | Chemical<br>Method | Q2 | Plasma | 4 |
| | Cardiac<br>troponin I | Venous | Elisa | Q2 | Serum | 4 |

## NOTES:

1. Sampling times: Pre-dose, End of Infusion, 0.5h, 1h, 2h, 4h, 8h, 24h, follow-up day 7-14

2. Sampling times: Pre-dose, 1h, 2h and 4h

3. Sampling times: Pre-dose, 2h, 4h and 24h

## 13.6. Appendix 6: Reporting Standards for Missing Data

## 13.6.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion (i.e. as specified in the protocol) was defined as a participant who has completed all phases of the study including the follow up visit and the last scheduled procedure</li> <li>Withdrawn subjects may be replaced in the study at the discretion of the sponsor.</li> <li>All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> </ul> |

## 13.6.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument:</li> <li>These data will be indicated by the use of a "blank" in subject listing displays. Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be missing data and should be displayed as such.</li> </ul> |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |
| Biomarkers | <ul> <li>Any values below the Lower Limit of Quantification (LLQ) will be assigned a value of ½ LLQ for display purposes in Figures and for computation of summary statistics. Any values above the Upper Limit of Quantification (ULQ) will be assigned to the ULQ for display purposes in Figures and for computation of summary statistics. If multiple LLQ and /or ULQ values are available per assay (for example if multiple runs with different standard curves are utilised) then the LLQ and/or ULQ value used for the above imputation shall be the minimum of the available LLQs and/or the maximum of the ULQs.</li> <li>If the number of LLQ (and/or ULQ) values is large for an individual biomarker then alternative analysis strategies may be required. "Large" is hard to define prospectively and may depend upon the dataset in question but a general rule of thumb is if &gt;30% of values are LLQ and/or ULQ. If "large" numbers of LLQ and/or ULQ values are observed methodologies to summarise and analyse the responses similar to those detailed in "Standards for the Handling of NQ impacted PK Parameters" (Respiratory DB and CPMS - 14th December 2009) may be employed. Any such methodology will be documented in the statistical contributions to the clinical study report.</li> </ul> |

For the derivation of the pulmonary wedge and venous (systemic) AngII / Ang(1-7) **ratios**, the following will apply:

| Flag | S | Numerator (ANGII) | | | |
|---|---|---|---|---|---|
| | | BLQ | Data | ALQ | Missing |
| (ANG1-7) | BLQ | (1/2 LLQ of ANGII) /<br>(1/2 LLQ of Ang(1-7)) | ANGII /<br>(1/2 LLQ of Ang(1-<br>7)) | (ULQ of ANGII) /<br>(1/2 LLQ of Ang(1-7)) | Missing |
| | Data | (1/2 LLQ of ANGII) /<br>Ang(1-7) | ANGII / Ang(1-7) | (ULQ of ANGII) /<br>Ang(1-7) | Missing |
| Denominator | ALQ | (1/2 LLQ of ANGII) /<br>(ULQ of Ang(1-7)) | ANGII /<br>(ULQ of Ang(1-7)) | (ULQ of ANGII) /<br>(ULQ of Ang(1-7)) | Missing |
| | Missing | Missing | Missing | Missing | Missing |
| LLQ | / ULQ = Lov | ver / Upper Limit of Quantificat | tion. BLQ / ALQ = Below / | Above Limit of Quantificati | on |

Note: The status of the numerator and denominator should be stored within derived datasets so they can be used in subsequent Summary Tables to display the amount of imputation necessary.

In addition, to support the PK/PD file to be generated (see Section 13.9.1), which will include the AngII/Ang(1-7) ratio, a variable will be included based on non-imputed data i.e., for this variable, the ratio will only be calculated if both AngII and Ang(1-7) have non-missing numeric values, otherwise the ratio will be set to missing.

#### 13.6.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse<br>Events | Missing or partial dates of AEs will not be allowed in this study. |
| Concomitant<br>Medications/<br>Medical<br>History | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> <li>The recorded partial date will be displayed in listings.</li> </ul> |

# 13.7. Appendix 7: Values of Potential Clinical Importance

## 13.7.1. Laboratory Values

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Cor | ncern Range |
| | | | Low Flag (< x) | High Flag (>x) |
| | | Male | | 0.54 |
| Hematocrit | Ratio of 1 | Female | | 0.54 |
| | | $\Delta$ from BL | ↓0.075 | |
| | a./I | Male | | 180 |
| Hemoglobin | g/L | Female | | 180 |
| | | $\Delta$ from BL | <b>↓25</b> | |
| Lymphocytes | x10 <sup>9</sup> / L | | 0.8 | |
| Neutrophil Count | x10 <sup>9</sup> / L | | 1.5 | |
| Platelet Count | x10 <sup>9</sup> / L | | 100 | 550 |
| While Blood Cell Count (WBC) | x10 <sup>9</sup> / L | | 3 | 20 |
| RBC Count | TI/L | | 0.93 x LLN | 1.07 x ULN |
| MCV | FL | | 0.25 x LLN | 2 x ULN |
| MCH | PG | | 0.85 x LLN | 1.1 x ULN |
| %Reticulocytes | % | | 0.5 x LLN | 5 x ULN |
| Monocytes | x10 <sup>9</sup> / L | | 0.25 x LLN | 2 x ULN |
| Eosinophils | x10 <sup>9</sup> / L | | 0 | 2 x ULN |
| Basophils | x10 <sup>9</sup> / L | | 0 | 5 x ULN |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Calcium | mmol/L | | 2 | 2.75 |
| Creatinine | mmol/L | | | ↑ 1.3 x ULN |
| Creatinine | mmol/L | $\Delta$ from BL | | ↑ 44.2 |
| Glucose | mmol/L | | 3 | 9 |
| Potassium | mmol/L | | 3 | 5.5 |
| Sodium | mmol/L | | 130 | 150 |
| BUN | mmol/L | | 0.7x | 1.6x |
| Direct Bilirubin | umol/L | | | 1.5x ULN |
| Total Protein | G/L | | | 1.25x |
| International normalized ratio | | On Warfarin | | 4 x |
| (INR) | | Not on Warfarin | | 1.5 x |
| Drothrombin time (DT) | | On Warfarin | | 4 x ULN |
| Prothrombin time (PT) | sec | Not on Warfarin | | 1.2 x ULN |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter Units Category Clinical Concern Range | | | | |
| | | | Low Flag (< x) | High Flag (>x) |
| PTT | Sec | On Heparin | | 4 x ULN |
| FII | Sec | Not on Heparin | | 1.2 x ULN |

| Liver Function | | | |
|--------------------|--------|----------|------------------------|
| Test Analyte | Units | Category | Clinical Concern Range |
| ALT/SGPT | U/L | High | ≥ 2x ULN |
| AST/SGOT | U/L | High | ≥ 2x ULN |
| AlkPhos | U/L | High | ≥ 2x ULN |
| T Bilirubin | µmol/L | High | ≥ 1.5xULN |
| | µmol/L | | 1.5xULN T. Bilirubin |
| T. Bilirubin + ALT | | High | + |
| | U/L | | ≥ 2x ULN ALT |
| Direct Bilirubin | | | 1.5 x ULN |

## 13.7.2. ECG

| ECG Parameter | Units | Clinical Concern Range | |
|----------------------------|-------|------------------------|-------|
| | | Lower | Upper |
| Absolute | | | |
| Absolute QTc Interval | msec | | ≥ 500 |
| Absolute PR Interval | msec | < 110 | > 220 |
| Absolute QRS Interval | msec | < 75 | > 110 |
| Change from Baseline | | | |
| Increase from Baseline QTc | msec | | > 60 |

## 13.7.3. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 90 | > 150 |
| Diastolic Blood Pressure | mmHg | < 50 | > 100 |
| Heart Rate | bpm | < 35 | > 130 |

| Vital Sign Parameter | Units | Clinical Concern Range | | | |
|---|---|---|---|---|---|
| (Change from Baseline) | | Decrease | | Increase | |
| | | Lower | Upper | Lower | Upper |
| Systolic Blood Pressure | mmHg | ≥ 20 | ≥ 40 | ≥ 20 | ≥ 40 |
| Diastolic Blood Pressure | mmHg | ≥ 10 | ≥ 20 | ≥ 10 | ≥ 20 |
| Heart Rate | bpm | ≥ 15 | ≥ 30 | ≥ 15 | ≥ 30 |

## 13.8. Appendix 8: Population Pharmacokinetic (PopPK) Analyses

## 13.8.1. Population Pharmacokinetic (PopPK) Dataset Specification

The PME compliant file structure is a space-delimited file with each row containing the following columns of information.

| Variable<br>short<br>name | Assessment description | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| С | Data Identifier | Integer | - | 0 |
| STUD | Protocol Number | Integer | - | 206246 |
| DRUG | Name of Drug | Integer | - | Maximum 10 characters (numeric or text). 2586881 |
| SUBJ | Subject identifier in study | Integer | - | Maximum 10 characters (numeric or text). Different identifier for each subject |
| CENT | Study centre identifier | Integer | - | |
| LABL | Indicator field describing the type of assessment in that record | Integer | See<br>footnot<br>es | See footnotes |
| AMT | Dose of<br>GSK2586881 | Decimal | Mg | Amount of drug given = Total<br>GSK2586881 dose (mg/kg)*WT<br>For dosing events: total dose of<br>GSK2586881 taken<br>For concentration events: 0 |
| INF | Infusion Time | Decimal | h | Time during which total dose infused. (Time at end of infusion – Time of start infusion) |
| RATE | Rate of Infusion | Decimal | Mg/h | Rate of infusion (AMT/INF) |
| DGRP | Treatment<br>Identifier | Decimal | - | DGRP = 0.1 for 0.1 mg/kg treatment<br>DGRP = 0.2 for 0.2 mg/kg treatment<br>DGRP = 0.4 for 0.4 mg/kg treatment<br>DGRP = 0.8 for 0.8 mg/kg treatment |
| PART | Study Part | Integer | - | 1=Study Period 1 |
| DAY | Study day | Integer | - | Maximum 10 characters (numeric or text) N= Day N, Actual Study Day |
| CTIM | Clock Time of Event | HH:MM:SS | - | Clock Time of Event |
| DATE | Date of Record | (DD/MM/YY<br>YY) | - | Date of Record |
| TRLD | Actual time relative to LAST dose | Decimal | Hours | When LABL = 1, 2, 3, or 4 TRLD is<br>Time (Hours) since start of LAST<br>infusion. For pre-dose sample,<br>TRLD=0 |
| DV | Dependent Variable | Decimal | pg/mL | When LABL=5, observed GSK2586881 concentration at time specified by TRLD. When LABL= 1, 2, 3 or 4 (dosing record), DV=0 |

| Variable<br>short<br>name | Assessment description | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| MDV | Missing Data<br>Variable | Integer | - | Either '0' if DV value present or 1 if DV value is non-quantifiable (NQ) or LABL = 1, 2, 3 or 4 |
| MDV1 | Missing data variable | Integer | - | Either '0' if LABL=5 or '1' if LABL= 1, 2, 3 or 4 |
| TYPE | F-Flag | Integer | - | If MDV1 = '1' then TYPE ='0', If DV value present (but not NQ) TYPE= '1' If DV value NQTYPE = '2' |
| LLQ | Lower Limit of quantification | Integer | pg/mL | Lower limit of quantification for specific analyte SMS dataset (PCLLQ) |
| CMT | Compartment data item | Integer | - | DOSE event: CMT=1, specifies the compartment into which DOSE is introduced. OBSERVATION event: CMT =1, specifies compartment from which observation is obtained. |
| AGE | Age | Decimal | Yrs | Integer. Age in years at time of screening rounded down to give age at last birthday. |
| WT | Weight | Decimal | Kg | Weight in kilograms at time of screening. |
| HT | Height | Decimal | Cm | Height in centimetres at time of screening. |
| SEX | Subject gender | Integer | - | Integer. One of the following - 1 = male 2 = female |
| ETHN | Subject ethnicity | Integer | - | Integer. Code as CRF |
| RACE | Subject race | Integer | - | Integer. Code as CRF |
| BMI | Body mass index | Decimal | kg/m^2 | body mass index calculated as weight divided by height squared |
| EVID | Event<br>Indentifcation data<br>item | Integer | - | Flag indicating whether LABL contains dosing admin info or drug concentration data. Valid values are - 1 – each dosing record for subject 0 - for all other records |

## Assessments captured in the LABL variable

| Label | Description | Units |
|---|---|---|
| 1 | Dosing records for 0.1 mg/Kg GSK2586881 | |
| 2 | Dosing records for 0.2 mg/Kg GSK2586881 | |
| 3 | Dosing records for 0.4 mg/Kg GSK2586881 | |
| 4 | Dosing records for 0.8 mg/Kg GSK2586881 | |
| 5 | Observed concentration record for GSK2586881 at time specified by TRLD; excludes NA, IS and NR, includes non-quantifiable (NQ) data | pg/mL |

## 13.9. Appendix 9: Pharmacokinetic / Pharmacodynamic Analyses

## 13.9.1. Pharmacokinetic / Pharmacodynamic Dataset Specification

## Specification for ANG II Venous (Systemic) [Proposed dataset name PKPDAIIV]

| Variable short name | Assessment description | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| С | Data Identifier | Integer | - | 0 |
| STUD | Protocol Number | Integer | - | 206246 |
| DRUG | Name of Drug | Integer | - | Maximum 10 characters (numeric or text). 2586881 |
| SUBJ | Subject identifier in study | Integer | - | Maximum 10 characters (numeric or text). Different identifier for each subject |
| CENT | Study centre identifier | Integer | - | |
| LABL | Indicator field describing the type of assessment in that record | Integer | See<br>footnotes | See footnotes |
| AMT | Dose of<br>GSK2586881 | Decimal | Mg | Amount of drug given = Total GSK2586881 dose (mg/kg) * WT. AMT=0 when LABL=0 For dosing events: total dose of GSK2586881 taken For concentration events: 0 |
| INF | Infusion Time | Decimal | h | Time during which total dose infused. (Time at end of infusion – Time of start infusion) |
| RATE | Rate of Infusion | Decimal | Mg/h | Rate of infusion (AMT/INF) |
| DGRP | Treatment Identifier | Decimal | - | DGRP=0.1 for 0.1 mg/kg treatment<br>DGRP=0.2 for 0.2 mg/kg treatment<br>DGRP=0.4 for 0.4 mg/kg treatment<br>DGRP=0.8 for 0.8 mg/kg treatment |
| PART | Study Part | Varchar | - | 1=Study Period 1 |
| DAY | Study day | Integer | - | Maximum 10 characters (numeric or text) N= Day N, Actual Study Day |
| CTIM | Clock time of Dose or measurement | HH:MM:SS | - | |
| DATE | Date of record | DD/MM/YYY | | |
| TRLD | Actual time relative to LAST dose | Decimal | Hours | When LABL = 1, 2, 3, or 4 TRLD is<br>Time (Hours) since start of LAST<br>infusion. For pre-dose sample,<br>TRLD=0 |
| BLII | Angll concentration record | Decimal | | Baseline value (pre-dose value) from venous (systemic) RAS sampling |

| Variable short name | Assessment description | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| DV | Angll concentration record | Decimal | | When LABL=6, observed AngII concentration at time specified by TRLD. When LABL= 1, 2, 3 or 4 (dosing record), DV=0, from venous (systemic) RAS sampling |
| MDV | Missing data variable | Integer | - | Either '0' if DV value present or 1 if DV is non-quantifiable (NQ) value or LABL= 1, 2, 3, or 4 |
| MDV1 | Missing data variable | Integer | - | '1' if LABL= 1, 2, 3 or 4<br>"0" when LABL=6 |
| TYPE | F-Flag | Integer | - | If MDV1= '1' then TYPE ='0', If DV value present (but not NQ) TYPE= '1' If DV value NQ TYPE = '2' |
| CMT | Compartment data item | Integer | - | DOSE event: CMT=1, specifies the compartment into which DOSE is introduced. OBSERVATION event: CMT=3 for DV (ANGII) observation event. |
| AGE | Age | Decimal | Yrs | Integer. Age in years at time of screening rounded down to give age at last birthday. |
| WT | Weight | Decimal | Kg | Weight in kilograms at time of screening. |
| HT | Height | Decimal | Cm | Height in centimetres at time of screening. |
| SEX | Subject gender | Integer | - | Integer. One of the following - 1 = male 2 = female |
| ETHN | Subject ethnicity | Integer | - | Integer. Code as CRF |
| RACE | Subject race | Integer | - | Integer. Code as CRF |
| BMI | Body mass index | Decimal | kg/m^2 | body mass index calculated as weight divided by height squared |
| EVID | Event Identification data item | Integer | - | Flag indicating whether LABL contains dosing admin info or drug concentration data. Valid values are - 1 – each dosing record for subject 0 - for all other records |

## Assessments captured in the LABL variable

| Label | Description | Units |
|---|---|---|
| 1 | Dosing records for 0.1 mg/Kg GSK2586881 | |
| 2 | Dosing records for 0.2 mg/Kg GSK2586881 | |
| 3 | Dosing records for 0.4 mg/Kg GSK2586881 | |
| 4 | Dosing records for 0.8 mg/Kg GSK2586881 | |
| 6 | Observed venous (systemic) sample ANGII record (concentration or ratio) at time specified by TRLD; excludes NA, IS and NR, includes non-quantifiable (NQ) data | |

## **Specification for ANG II Pulmonary Wedge [proposed dataset name PKPDAIIP]**

| Variable | Assessment | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| short name | description Data Identifier | Intogor | <u> </u> | 0 |
| STUD | Protocol Number | Integer | <del>-</del><br> - | 206246 |
| DRUG | Name of Drug | Integer<br>Integer | - | Maximum 10 characters (numeric or text). 2586881 |
| SUBJ | Subject identifier in study | Integer | - | Maximum 10 characters (numeric or text). Different identifier for each subject |
| CENT | Study centre identifier | Integer | - | |
| LABL | Indicator field describing the type of assessment in that record | Integer | See<br>footnotes | See footnotes |
| AMT | Dose of<br>GSK2586881 | Decimal | Mg | Amount of drug given = Total GSK2586881 dose (mg/kg) * WT. AMT=0 when LABL=0 For dosing events: total dose of GSK2586881 taken For concentration events: 0 |
| INF | Infusion Time | Decimal | h | Time during which total dose infused. (Time at end of infusion – Time of start infusion) |
| RATE | Rate of Infusion | Decimal | Mg/h | Rate of infusion (AMT/INF) |
| DGRP | Treatment Identifier | Decimal | - | DGRP=0.1 for 0.1 mg/kg treatment<br>DGRP=0.2 for 0.2 mg/kg treatment<br>DGRP=0.4 for 0.4 mg/kg treatment<br>DGRP=0.8 for 0.8 mg/kg treatment |
| PART | Study Part | Varchar | - | 1=Study Period 1 |
| DAY | Study day | Integer | - | Maximum 10 characters (numeric or text) N= Day N, Actual Study Day |
| СТІМ | Clock time of Dose or measurement | HH:MM:SS | - | |
| DATE | Date of record | DD/MM/YYY | | |
| TRLD | Actual time relative | Decimal | Hours | When LABL = 1, 2, 3, or 4 TRLD is |

| Variable short name | Assessment description | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| | to LAST dose | | | Time (Hours) since start of LAST infusion. For pre-dose sample, TRLD=0 |
| BLII | Angll concentration record | Decimal | | Baseline value (pre-dose value) from pulmonary wedge RAS sampling |
| DV | Angll concentration record | Decimal | | When LABL=11, observed AngII concentration at time specified by TRLD. When LABL= 1, 2, 3 or 4 (dosing record), DV=0, from pulmonary wedge RAS sampling |
| MDV | Missing data variable | Integer | - | Either '0' if DV value present or 1 if DV is non-quantifiable (NQ) value or LABL= 1, 2, 3, or 4 |
| MDV1 | Missing data variable | Integer | - | '1' if LABL= 1, 2, 3 or 4<br>"0" when LABL=11 |
| TYPE | F-Flag | Integer | - | If MDV1= '1' then TYPE ='0', If DV value present (but not NQ) TYPE= '1' If DV value NQ TYPE = '2' |
| CMT | Compartment data item | Integer | - | DOSE event: CMT=1, specifies the compartment into which DOSE is introduced. OBSERVATION event: CMT=3 for DV (ANGII) observation event. |
| AGE | Age | Decimal | Yrs | Integer. Age in years at time of screening rounded down to give age at last birthday. |
| WT | Weight | Decimal | Kg | Weight in kilograms at time of screening. |
| HT | Height | Decimal | Cm | Height in centimetres at time of screening. |
| SEX | Subject gender | Integer | - | Integer. One of the following - 1 = male 2 = female |
| ETHN | Subject ethnicity | Integer | - | Integer. Code as CRF |
| RACE | Subject race | Integer | - | Integer. Code as CRF |
| BMI | Body mass index | Decimal | kg/m^2 | body mass index calculated as weight divided by height squared |
| EVID | Event Identification data item | Integer | - | Flag indicating whether LABL contains dosing admin info or drug concentration data. Valid values are - 1 – each dosing record for subject 0 - for all other records |

## Assessments captured in the LABL variable

| Label | Description | Units |
|---|---|---|
| 1 | Dosing records for 0.1 mg/Kg GSK2586881 | |
| 2 | Dosing records for 0.2 mg/Kg GSK2586881 | |
| 3 | Dosing records for 0.4 mg/Kg GSK2586881 | |
| 4 | Dosing records for 0.8 mg/Kg GSK2586881 | |
| 11 | Observed pulmonary wedge sample ANGII record (concentration or ratio) at time specified by TRLD; excludes NA, IS and NR, includes non-quantifiable (NQ) data | |

## Specification for ANG(1-5) Venous (Systemic) [proposed dataset name PKPDA15V]

| Variable short name | Assessment | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| C | description Data Identifier | Intogor | <del> </del> | 0 |
| STUD | Protocol Number | Integer<br>Integer | -<br> _ | 206246 |
| DRUG | Name of Drug | Integer | - | Maximum 10 characters (numeric or text). 2586881 |
| SUBJ | Subject identifier in study | Integer | - | Maximum 10 characters (numeric or text). Different identifier for each subject |
| CENT | Study centre identifier | Integer | - | |
| LABL | Indicator field describing the type of assessment in that record | Integer | See<br>footnotes | See footnotes |
| AMT | Dose of<br>GSK2586881 | Decimal | Mg | Amount of drug given = Total GSK2586881 dose (mg/kg) * WT. AMT=0 when LABL=0 For dosing events: total dose of GSK2586881 taken For concentration events: 0 |
| INF | Infusion Time | Decimal | Н | Time during which total dose infused. (Time at end of infusion – Time of start infusion) |
| RATE | Rate of Infusion | Decimal | Mg/h | Rate of infusion (AMT/INF) |
| DGRP | Treatment Identifier | Decimal | - | DGRP=0.1 for 0.1 mg/kg treatment<br>DGRP=0.2 for 0.2 mg/kg treatment<br>DGRP=0.4 for 0.4 mg/kg treatment<br>DGRP=0.8 for 0.8 mg/kg treatment |
| PART | Study Part | Varchar | - | 1=Study Period 1 |
| DAY | Study day | Integer | - | Maximum 10 characters (numeric or text) N= Day N, Actual Study Day |
| CTIM | Clock time of Dose or measurement | HH:MM:SS | - | |
| DATE | Date of record | DD/MM/YYY | | |
| TRLD | Actual time relative | Decimal | Hours | When LABL = 1, 2, 3, or 4 TRLD is |

| Variable short name | Assessment description | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| | to LAST dose | | | Time (Hours) since start of LAST infusion. For pre-dose sample, TRLD=0 |
| BL15 | Ang1-5 concentration record | Decimal | | Baseline value, from venous (systemic) RAS sampling |
| DV | Angl1-5 concentration record | Decimal | | When LABL=7, observed Ang1-5 concentration at time specified by TRLD. When LABL= 1, 2, 3 or 4 (dosing record), DV=0, from venous (systemic) RAS sampling |
| MDV | Missing data variable | Integer | - | Either '0' if DV value present or 1 if DV is non-quantifiable (NQ) value or LABL=1, 2, 3 or 4 |
| MDV1 | Missing data variable | Integer | - | '1' if LABL=1, 2, 3 or 4<br>"0" when LABL=7 |
| TYPE | F-Flag | Integer | - | If MDV1= '1' then TYPE ='0', If DV value present (but not NQ) TYPE= '1' If DV value NQ TYPE = '2' |
| CMT | Compartment data item | Integer | - | DOSE event: CMT=1, specifies the compartment into which DOSE is introduced. OBSERVATION event CMT=4 for ANG1-5 observation event. |
| AGE | Age | Decimal | Yrs | Integer. Age in years at time of screening rounded down to give age at last birthday. |
| WT | Weight | Decimal | Kg | Weight in kilograms at time of screening. |
| HT | Height | Decimal | Cm | Height in centimetres at time of screening. |
| SEX | Subject gender | Integer | - | Integer. One of the following - 1 = male 2 = female |
| ETHN | Subject ethnicity | Integer | - | Integer. Code as CRF |
| RACE | Subject race | Integer | - | Integer. Code as CRF |
| BMI | Body mass index | Decimal | kg/m^2 | body mass index calculated as weight divided by height squared |
| EVID | Event Identification data item | Integer | - | Flag indicating whether LABL contains dosing admin info or drug concentration data. Valid values are - 1 – each dosing record for subject 0 - for all other records |

## Assessments captured in the LABL variable

| Label | Description | Units |
|---|---|---|
| 1 | Dosing records for 0.1 mg/Kg GSK2586881 | |
| 2 | Dosing records for 0.2 mg/Kg GSK2586881 | |
| 3 | Dosing records for 0.4 mg/Kg GSK2586881 | |
| 4 | Dosing records for 0.8 mg/Kg GSK2586881 | |
| 7 | Observed venous (systemic) sampling ANG15 record (concentration or ratio) at time specified by TRLD; excludes NA, IS and NR, includes non-quantifiable (NQ) data | |

## Specification for ANG(1-5) Pulmonary Wedge [proposed dataset name PKPDA15P]

| Variable | Assessment | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| short name | description | | | |
| С | Data Identifier | Integer | - | 0 |
| STUD | Protocol Number | Integer | - | 206246 |
| DRUG | Name of Drug | Integer | - | Maximum 10 characters (numeric or text). 2586881 |
| SUBJ | Subject identifier in study | Integer | - | Maximum 10 characters (numeric or text). Different identifier for each subject |
| CENT | Study centre identifier | Integer | - | |
| LABL | Indicator field describing the type of assessment in that record | Integer | See<br>footnotes | See footnotes |
| AMT | Dose of<br>GSK2586881 | Decimal | Mg | Amount of drug given = Total GSK2586881 dose (mg/kg) * WT. AMT=0 when LABL=0 For dosing events: total dose of GSK2586881 taken For concentration events: 0 |
| INF | Infusion Time | Decimal | Н | Time during which total dose infused. (Time at end of infusion – Time of start infusion) |
| RATE | Rate of Infusion | Decimal | Mg/h | Rate of infusion (AMT/INF) |
| DGRP | Treatment Identifier | Decimal | - | DGRP=0.1 for 0.1 mg/kg treatment<br>DGRP=0.2 for 0.2 mg/kg treatment<br>DGRP=0.4 for 0.4 mg/kg treatment<br>DGRP=0.8 for 0.8 mg/kg treatment |
| PART | Study Part | Varchar | - | 1=Study Period 1 |
| DAY | Study day | Integer | - | Maximum 10 characters (numeric or text) N= Day N, Actual Study Day |
| CTIM | Clock time of Dose or measurement | HH:MM:SS | - | |
| DATE | Date of record | DD/MM/YYY | | |

| Variable short name | Assessment description | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| TRLD | Actual time relative to LAST dose | Decimal | Hours | When LABL = 1, 2, 3, or 4 TRLD is<br>Time (Hours) since start of LAST<br>infusion. For pre-dose sample,<br>TRLD=0 |
| BL15 | Ang1-5 concentration record | Decimal | | Baseline value, from pulmonary wedge RAS sampling |
| DV | Angl1-5<br>concentration<br>record | Decimal | | When LABL=12, observed Ang1-5 concentration at time specified by TRLD. When LABL= 1, 2, 3 or 4 (dosing record), DV=0, from pulmonary wedge RAS sampling |
| MDV | Missing data variable | Integer | - | Either '0' if DV value present or 1 if DV is non-quantifiable (NQ) value or LABL=1, 2, 3 or 4 |
| MDV1 | Missing data variable | Integer | - | '1' if LABL=1, 2, 3 or 4<br>"0" when LABL=12 |
| TYPE | F-Flag | Integer | - | If MDV1= '1' then TYPE ='0', If DV value present (but not NQ) TYPE= '1' If DV value NQ TYPE = '2' |
| CMT | Compartment data item | Integer | - | DOSE event: CMT=1, specifies the compartment into which DOSE is introduced. OBSERVATION event CMT=4 for ANG1-5 observation event. |
| AGE | Age | Decimal | Yrs | Integer. Age in years at time of screening rounded down to give age at last birthday. |
| WT | Weight | Decimal | Kg | Weight in kilograms at time of screening. |
| HT | Height | Decimal | Cm | Height in centimetres at time of screening. |
| SEX | Subject gender | Integer | - | Integer. One of the following - 1 = male 2 = female |
| ETHN | Subject ethnicity | Integer | - | Integer. Code as CRF |
| RACE | Subject race | Integer | - | Integer. Code as CRF |
| BMI | Body mass index | Decimal | kg/m^2 | body mass index calculated as weight divided by height squared |
| EVID | Event Identification data item | Integer | - | Flag indicating whether LABL contains dosing admin info or drug concentration data. Valid values are - 1 – each dosing record for subject 0 - for all other records |

## Assessments captured in the LABL variable

| Label | Description | Units |
|---|---|---|
| 1 | Dosing records for 0.1 mg/Kg GSK2586881 | |
| 2 | Dosing records for 0.2 mg/Kg GSK2586881 | |
| 3 | Dosing records for 0.4 mg/Kg GSK2586881 | |
| 4 | Dosing records for 0.8 mg/Kg GSK2586881 | |
| 12 | Observed pulmonary wedge sampling ANG15 record (concentration or ratio) at time specified by TRLD; excludes NA, IS and NR, includes non-quantifiable (NQ) data | |

## Specification for ANG(1-7) Venous (Systemic) [proposed dataset name PKPDA17V]

| Variable short name | Assessment description | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| С | Data Identifier | Integer | - | 0 |
| STUD | Protocol Number | Integer | - | 206246 |
| DRUG | Name of Drug | Integer | - | Maximum 10 characters (numeric or text). 2586881 |
| SUBJ | Subject identifier in study | Integer | - | Maximum 10 characters (numeric or text). Different identifier for each subject |
| CENT | Study centre identifier | Integer | - | |
| LABL | Indicator field describing the type of assessment in that record | Integer | See<br>footnotes | See footnotes |
| AMT | Dose of<br>GSK2586881 | Decimal | Mg | Amount of drug given = Total GSK2586881 dose (mg/kg) * WT. AMT=0 when LABL=0 For dosing events: total dose of GSK2586881 taken For concentration events: 0 |
| INF | Infusion Time | Decimal | Н | Time during which total dose infused. (Time at end of infusion – Time of start infusion) |
| RATE | Rate of Infusion | Decimal | Mg/h | Rate of infusion (AMT/INF) |
| DGRP | Treatment Identifier | Decimal | - | DGRP=0.1 for 0.1 mg/kg treatment<br>DGRP=0.2 for 0.2 mg/kg treatment<br>DGRP=0.4 for 0.4 mg/kg treatment<br>DGRP=0.8 for 0.8 mg/kg treatment |
| PART | Study Part | Varchar | - | 1=Study Period 1 |
| DAY | Study day | Integer | - | Maximum 10 characters (numeric or text) N= Day N, Actual Study Day |
| CTIM | Clock time of Dose or measurement | HH:MM:SS | - | |
| DATE | Date of record | DD/MM/YYY | | |
| TRLD | Actual time relative | Decimal | Hours | When LABL = 1, 2, 3, or 4 TRLD is |

| Variable short name | Assessment description | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| | to LAST dose | | | Time (Hours) since start of LAST infusion. For pre-dose sample, TRLD=0 |
| BL17 | Ang1-7 concentration record | Decimal | | Baseline value, from venous (systemic) RAS sampling |
| DV | Ang1-7 concentration record | Decimal | | When LABL=8, observed Ang1-7 concentration at time specified by TRLD. When LABL= 1, 2, 3 or 4 (dosing record), DV=0, from venous (systemic) RAS sampling |
| MDV | Missing data variable | Integer | - | Either '0' if DV value present or 1 if DV is non-quantifiable (NQ) value or LABL=1, 2, 3 or 4 |
| MDV1 | Missing data variable | Integer | - | '1' if LABL=1, 2, 3 or 4<br>"0" when LABL=8 |
| TYPE | F-Flag | Integer | - | If MDV1= '1' then TYPE ='0', If ANG1-7 value present (but not NQ) TYPE= '1' If ANG1-7 value NQ TYPE = '2' |
| CMT | Compartment data item | Integer | - | DOSE event: CMT=1, specifies the compartment into which DOSE is introduced. OBSERVATION event: CMT=5 for ANG1-7 observation event. |
| AGE | Age | Decimal | Yrs | Integer. Age in years at time of screening rounded down to give age at last birthday. |
| WT | Weight | Decimal | Kg | Weight in kilograms at time of screening. |
| HT | Height | Decimal | Cm | Height in centimetres at time of screening. |
| SEX | Subject gender | Integer | - | Integer. One of the following - 1 = male 2 = female |
| ETHN | Subject ethnicity | Integer | - | Integer. Code as CRF |
| RACE | Subject race | Integer | - | Integer. Code as CRF |
| BMI | Body mass index | Decimal | kg/m^2 | body mass index calculated as weight divided by height squared |
| EVID | Event Identification data item | Integer | - | Flag indicating whether LABL contains dosing admin info or drug concentration data. Valid values are - 1 – each dosing record for subject 0 - for all other records |

## Assessments captured in the LABL variable

| Label | Description | Units |
|---|---|---|
| 1 | Dosing records for 0.1 mg/Kg GSK2586881 | |
| 2 | Dosing records for 0.2 mg/Kg GSK2586881 | |
| 3 | Dosing records for 0.4 mg/Kg GSK2586881 | |
| 4 | Dosing records for 0.8 mg/Kg GSK2586881 | |
| 8 | Observed venous (systemic) sampling ANG17 record (concentration or ratio) at time specified by TRLD; excludes NA, IS and NR, includes non-quantifiable (NQ) data | |

## Specification for ANG(1-7) Pulmonary Wedge [proposed dataset name PKPDA17P]

| Variable short name | Assessment description | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| С | Data Identifier | Integer | - | 0 |
| STUD | Protocol Number | Integer | - | 206246 |
| DRUG | Name of Drug | Integer | - | Maximum 10 characters (numeric or text). 2586881 |
| SUBJ | Subject identifier in study | Integer | - | Maximum 10 characters (numeric or text). Different identifier for each subject |
| CENT | Study centre identifier | Integer | - | |
| LABL | Indicator field describing the type of assessment in that record | Integer | See<br>footnotes | See footnotes |
| AMT | Dose of<br>GSK2586881 | Decimal | Mg | Amount of drug given = Total GSK2586881 dose (mg/kg) * WT. AMT=0 when LABL=0 For dosing events: total dose of GSK2586881 taken For concentration events: 0 |
| INF | Infusion Time | Decimal | Н | Time during which total dose infused. (Time at end of infusion – Time of start infusion) |
| RATE | Rate of Infusion | Decimal | Mg/h | Rate of infusion (AMT/INF) |
| DGRP | Treatment Identifier | Decimal | - | DGRP=0.1 for 0.1 mg/kg treatment<br>DGRP=0.2 for 0.2 mg/kg treatment<br>DGRP=0.4 for 0.4 mg/kg treatment<br>DGRP=0.8 for 0.8 mg/kg treatment |
| PART | Study Part | Varchar | - | 1=Study Period 1 |
| DAY | Study day | Integer | - | Maximum 10 characters (numeric or text) N= Day N, Actual Study Day |
| CTIM | Clock time of Dose or measurement | HH:MM:SS | - | |
| DATE | Date of record | DD/MM/YYY | | |
| TRLD | Actual time relative | Decimal | Hours | When LABL = 1, 2, 3, or 4 TRLD is |

| Variable short name | Assessment description | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| | to LAST dose | | | Time (Hours) since start of LAST infusion. For pre-dose sample, TRLD=0 |
| BL17 | Ang1-7 concentration record | Decimal | | Baseline value, from pulmonary wedge RAS sampling |
| DV | Ang1-7 concentration record | Decimal | | When LABL=13, observed Ang1-7 concentration at time specified by TRLD. When LABL= 1, 2, 3 or 4 (dosing record), DV=0, from pulmonary wedge RAS sampling |
| MDV | Missing data variable | Integer | - | Either '0' if DV value present or 1 if DV is non-quantifiable (NQ) value or LABL=1, 2, 3 or 4 |
| MDV1 | Missing data variable | Integer | - | '1' if LABL=1, 2, 3 or 4<br>"0" when LABL=13 |
| TYPE | F-Flag | Integer | - | If MDV1= '1' then TYPE ='0', If ANG1-7 value present (but not NQ) TYPE= '1' If ANG1-7 value NQTYPE = '2' |
| CMT | Compartment data item | Integer | - | DOSE event: CMT=1, specifies the compartment into which DOSE is introduced. OBSERVATION event: CMT=5 for ANG1-7 observation event. |
| AGE | Age | Decimal | Yrs | Integer. Age in years at time of screening rounded down to give age at last birthday. |
| WT | Weight | Decimal | Kg | Weight in kilograms at time of screening. |
| HT | Height | Decimal | Cm | Height in centimetres at time of screening. |
| SEX | Subject gender | Integer | - | Integer. One of the following -<br>1 = male<br>2 = female |
| ETHN | Subject ethnicity | Integer | - | Integer. Code as CRF |
| RACE | Subject race | Integer | - | Integer. Code as CRF |
| BMI | Body mass index | Decimal | kg/m^2 | body mass index calculated as weight divided by height squared |
| EVID | Event Identification data item | Integer | - | Flag indicating whether LABL contains dosing admin info or drug concentration data. Valid values are - 1 – each dosing record for subject 0 - for all other records |

## Assessments captured in the LABL variable

| Label | Description | Units |
|---|---|---|
| 1 | Dosing records for 0.1 mg/Kg GSK2586881 | |
| 2 | Dosing records for 0.2 mg/Kg GSK2586881 | |
| 3 | Dosing records for 0.4 mg/Kg GSK2586881 | |
| 4 | Dosing records for 0.8 mg/Kg GSK2586881 | |
| 13 | Observed pulmonary wedge sampling ANG17 record (concentration or ratio) at time specified by TRLD; excludes NA, IS and NR, includes non-quantifiable (NQ) data | |

# Specification for ANGII/ANG(1-7) Venous (Systemic) [proposed dataset name PKPDARTV]

| Variable short name | Assessment description | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| С | Data Identifier | Integer | - | 0 |
| STUD | Protocol Number | Integer | - | 206246 |
| DRUG | Name of Drug | Integer | - | Maximum 10 characters (numeric or text). 2586881 |
| SUBJ | Subject identifier in study | Integer | - | Maximum 10 characters (numeric or text). Different identifier for each subject |
| CENT | Study centre identifier | Integer | - | |
| LABL | Indicator field describing the type of assessment in that record | Integer | See<br>footnotes | See footnotes |
| AMT | Dose of<br>GSK2586881 | Decimal | Mg | Amount of drug given = Total GSK2586881 dose (mg/kg) * WT. AMT=0 when LABL=0 For dosing events: total dose of GSK2586881 taken For concentration events: 0 |
| INF | Infusion Time | Decimal | Н | Time during which total dose infused. (Time at end of infusion – Time of start infusion) |
| RATE | Rate of Infusion | Decimal | Mg/h | Rate of infusion (AMT/INF) |
| DGRP | Treatment Identifier | Decimal | - | DGRP=0.1 for 0.1 mg/kg treatment<br>DGRP=0.2 for 0.2 mg/kg treatment<br>DGRP=0.4 for 0.4 mg/kg treatment<br>DGRP=0.8 for 0.8 mg/kg treatment |
| PART | Study Part | Varchar | - | 1=Study Period 1 |
| DAY | Study day | Integer | - | Maximum 10 characters (numeric or text) N= Day N, Actual Study Day |
| CTIM | Clock time of Dose or measurement | HH:MM:SS | - | |

| Variable short name | Assessment description | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| DATE | Date of record | DD/MM/YYY | | |
| TRLD | Actual time relative to LAST dose | Decimal | Hours | When LABL = 1, 2, 3, or 4 TRLD is<br>Time (Hours) since start of LAST<br>infusion. For pre-dose sample,<br>TRLD=0 |
| BLRT | AngII/Ang1-7 ratio concentration record | Decimal | | Baseline value, from venous (systemic) RAS sampling Refer to Section 13.6.2 for details of data to include. |
| DV | AngII/Ang1-7 ratio concentration record | Decimal | | When LABL=10, observed AngII/Ang1-7 ratio at time specified by TRLD. When LABL= 1, 2, 3 or 4 (dosing record), DV=0, from venous (systemic) RAS sampling Refer to Section 13.6.2 for details of data to include. |
| MDV | Missing data variable | Integer | - | Either '0' if DV value present or 1 if DV is non-quantifiable (NQ) value or missing value or LABL=1, 2, 3 or 4 |
| MDV1 | Missing data variable | Integer | - | '1' if LABL=1, 2, 3 or 4<br>"0" when LABL=10 |
| TYPE | F-Flag | Integer | - | If MDV1= '1' then TYPE ='0', If ANGII/ANG1-7 value present (but not NQ) TYPE= '1' If ANGII/ANG1-7 value NQ (or missing) TYPE = '2' |
| CMT | Compartment data item | Integer | - | DOSE event: CMT=1, specifies the compartment into which DOSE is introduced. OBSERVATION event: CMT=6 for ANGII/ANG1-7 observation event. |
| AGE | Age | Decimal | Yrs | Integer. Age in years at time of screening rounded down to give age at last birthday. |
| WT | Weight | Decimal | Kg | Weight in kilograms at time of screening. |
| HT | Height | Decimal | Cm | Height in centimetres at time of screening. |
| SEX | Subject gender | Integer | - | Integer. One of the following -<br>1 = male<br>2 = female |
| ETHN | Subject ethnicity | Integer | - | Integer. Code as CRF |
| RACE | Subject race | Integer | - | Integer. Code as CRF |
| BMI | Body mass index | Decimal | kg/m^2 | body mass index calculated as |

| Variable short name | Assessment description | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| | | | | weight divided by height squared |
| EVID | Event Identification data item | Integer | - | Flag indicating whether LABL contains dosing admin info or drug concentration data. Valid values are - 1 – each dosing record for subject 0 - for all other records |

## Assessments captured in the LABL variable

| Label | Description | Units |
|---|---|---|
| 1 | Dosing records for 0.1 mg/Kg GSK2586881 | |
| 2 | Dosing records for 0.2 mg/Kg GSK2586881 | |
| 3 | Dosing records for 0.4 mg/Kg GSK2586881 | |
| 4 | Dosing records for 0.8 mg/Kg GSK2586881 | |
| 10 | Observed venous (systemic) sampling ANGII/ANG17 record (ratio) at time specified by TRLD; excludes NA, IS and NR, includes non-quantifiable (NQ) data | |

# Specification for ANGII/ANG(1-7) Pulmonary Wedge [proposed dataset name PKPDARTP]

| Variable short name | Assessment description | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| С | Data Identifier | Integer | - | 0 |
| STUD | Protocol Number | Integer | - | 206246 |
| DRUG | Name of Drug | Integer | - | Maximum 10 characters (numeric or text). 2586881 |
| SUBJ | Subject identifier in study | Integer | - | Maximum 10 characters (numeric or text). Different identifier for each subject |
| CENT | Study centre identifier | Integer | - | |
| LABL | Indicator field describing the type of assessment in that record | Integer | See<br>footnotes | See footnotes |
| AMT | Dose of<br>GSK2586881 | Decimal | Mg | Amount of drug given = Total GSK2586881 dose (mg/kg) * WT. AMT=0 when LABL=0 For dosing events: total dose of GSK2586881 taken For concentration events: 0 |
| INF | Infusion Time | Decimal | Н | Time during which total dose infused. (Time at end of infusion – Time of start infusion) |
| RATE | Rate of Infusion | Decimal | Mg/h | Rate of infusion (AMT/INF) |

| Variable short name | Assessment description | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| DGRP | Treatment Identifier | Decimal | - | DGRP=0.1 for 0.1 mg/kg treatment<br>DGRP=0.2 for 0.2 mg/kg treatment<br>DGRP=0.4 for 0.4 mg/kg treatment<br>DGRP=0.8 for 0.8 mg/kg treatment |
| PART | Study Part | Varchar | - | 1=Study Period 1 |
| DAY | Study day | Integer | - | Maximum 10 characters (numeric or text) N= Day N, Actual Study Day |
| CTIM | Clock time of Dose or measurement | HH:MM:SS | - | |
| DATE | Date of record | DD/MM/YYY | | |
| TRLD | Actual time relative to LAST dose | Decimal | Hours | When LABL = 1, 2, 3, or 4 TRLD is<br>Time (Hours) since start of LAST<br>infusion. For pre-dose sample,<br>TRLD=0 |
| BLRT | AngII/Ang1-7 ratio concentration record | Decimal | | Baseline value, from pulmonary wedge RAS sampling Refer to Section 13.6.2 for details of data to include. |
| DV | AngII/Ang1-7 ratio concentration record | Decimal | | When LABL=14, observed AngIl/Ang1-7 ratio at time specified by TRLD. When LABL= 1, 2, 3 or 4 (dosing record), DV=0, from pulmonary wedge RAS sampling Refer to Section 13.6.2 for details of data to include. |
| MDV | Missing data variable | Integer | - | Either '0' if DV value present or 1 if DV is non-quantifiable (NQ) value or missing value or LABL=1, 2, 3 or 4 |
| MDV1 | Missing data variable | Integer | - | '1' if LABL=1, 2, 3 or 4<br>"0" when LABL=14 |
| TYPE | F-Flag | Integer | - | If MDV1= '1' then TYPE ='0', If ANGII/ANG1-7 value present (but not NQ) TYPE= '1' If ANGII/ANG1-7 value NQ (or missing) TYPE = '2' |
| CMT | Compartment data item | Integer | - | DOSE event: CMT=1, specifies the compartment into which DOSE is introduced. OBSERVATION event: CMT=6 for ANGII/ ANG1-7 observation event. |
| AGE | Age | Decimal | Yrs | Integer. Age in years at time of screening rounded down to give age at last birthday. |
| WT | Weight | Decimal | Kg | Weight in kilograms at time of |

| Variable short name | Assessment description | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| | | | | screening. |
| HT | Height | Decimal | Cm | Height in centimetres at time of screening. |
| SEX | Subject gender | Integer | - | Integer. One of the following -<br>1 = male<br>2 = female |
| ETHN | Subject ethnicity | Integer | - | Integer. Code as CRF |
| RACE | Subject race | Integer | - | Integer. Code as CRF |
| BMI | Body mass index | Decimal | kg/m^2 | body mass index calculated as weight divided by height squared |
| EVID | Event Identification data item | Integer | - | Flag indicating whether LABL contains dosing admin info or drug concentration data. Valid values are - 1 – each dosing record for subject 0 - for all other records |

## Assessments captured in the LABL variable

| Label | Description | Units |
|---|---|---|
| 1 | Dosing records for 0.1 mg/Kg GSK2586881 | |
| 2 | Dosing records for 0.2 mg/Kg GSK2586881 | |
| 3 | Dosing records for 0.4 mg/Kg GSK2586881 | |
| 4 | Dosing records for 0.8 mg/Kg GSK2586881 | |
| 14 | Observed pulmonary wedge sampling ANGII/ANG17 record (ratio) at time specified by TRLD; excludes NA, IS and NR, includes non-quantifiable (NQ) data | |

## **Specification for PVR/CO/mPAP/CI**

The PME compliant file structure is a space-delimited file with each row containing the following columns of information. Data from all treatments will be included.

| Variable short name | Assessment description | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| С | Data Identifier | Integer | - | 0 |
| STUD | Protocol Number | Integer | - | 206246 |
| DRUG | Name of Drug | Integer | - | Maximum 10 characters (numeric or text). 2586881 |
| SUBJ | Subject identifier in study | Integer | - | Maximum 10 characters (numeric or text). Different identifier for each subject |
| CENT | Study centre identifier | Integer | - | |
| LABL | Indicator field describing the type of assessment in | Integer | See<br>footnotes | See footnotes |

| Variable | Assessment | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| short name | description | | | |
| | that record | | | |
| AMT | Dose of<br>GSK2586881 | Decimal | Mg | Amount of drug given = Total GSK2586881 dose (mg/kg) * WT. AMT=0 when LABL=0 For dosing events: total dose of GSK2586881 taken For concentration events: 0 |
| INF | Infusion Time | Decimal | h | Time during which total dose infused. (Time at end of infusion – Time of start infusion) |
| RATE | Rate of Infusion | Decimal | Mg/h | Rate of infusion (AMT/INF) |
| DGRP | Treatment Identifier | Decimal | - | DGRP=0.1 for 0.1 mg/kg treatment<br>DGRP=0.2 for 0.2 mg/kg treatment<br>DGRP=0.4 for 0.4 mg/kg treatment<br>DGRP=0.8 for 0.8 mg/kg treatment |
| PART | Study Part | Varchar | - | 1=Study Period 1 |
| DAY | Study day | Integer | - | Maximum 10 characters (numeric or text) N= Day N, Actual Study Day |
| CTIM | Clock time of Dose or measurement | HH:MM:SS | - | |
| DATE | Date of record | DD/MM/YYY | | |
| TRLD | Actual time relative to LAST dose | Decimal | Hours | When LABL = 1, 2, 3, or 4 TRLD is<br>Time (Hours) since start of LAST<br>infusion. For pre-dose sample,<br>TRLD=0 |
| BLPVR | PVR | Decimal | mmHg | Baseline Value |
| PVR | PVR | Decimal | mmHg | When LABL=9, PVR at time specified by TRLD. When LABL= 1, 2, 3 or 4 (dosing record), PVR=0 |
| PVRFLD | PVR ratio to baseline (fold change) | Decimal | - | When LABL=9, PVRFLD fold change at time specified by TRLD. When LABL= 1, 2, 3 or 4 (dosing record), PVRFLD=0 |
| PVRCHG | PVR change from baseline | Decimal | mmHg | When LABL=9, PVRCHG at time specified by TRLD. When LABL= 1, 2, 3 or 4 (dosing record), PVRCHG=0 |
| BLCO | Cardiac Output | Decimal | L/min | Baseline Value |
| CO | Cardiac Output | Decimal | L/min | When LABL=9, CO at time specified by TRLD. When LABL= 1, 2, 3 or 4 (dosing record), DV=0 CO=0 |
| COFLD | Cardiac Output<br>ratio to baseline<br>(fold change) | Decimal | - | When LABL=9, COFLD fold change at time specified by TRLD. When LABL= 1, 2, 3 or 4 (dosing record), DV=0 COFLD=0 |
| COCHG | Cardiac Output | Decimal | L/min | When LABL=9, COCHG at time |

| Variable short name | Assessment description | Format | Unit | Valid Values / Format |
|---|---|---|---|---|
| | change from baseline | | | specified by TRLD. When LABL=<br>1, 2, 3 or 4 (dosing record), DV=0<br>COCHG=0 |
| BLCI | Cardiac Index | Decimal | L/min/m2 | Baseline Value |
| CI | Cardiac Index | Decimal | L/min/m2 | When LABL=9, CI at time specified by TRLD. When LABL= 1, 2, 3 or 4 (dosing record), DV=0 CI=0 |
| CIFLD | Cardiac Index ratio<br>to baseline (fold<br>change) | Decimal | - | When LABL=9, CIFLD fold change at time specified by TRLD. When LABL=1, 2, 3 or 4 (dosing record), DV=0 CIFLD=0. |
| CICHG | Cardiac Index<br>change from<br>baseline | Decimal | L/min/m2 | When LABL=9, CICHG at time specified by TRLD. When LABL=1, 2, 3 or 4 (dosing record), DV=0 CICHG=0. |
| BLMPAP | mPAP | Decimal | mmHg | Baseline Value |
| MPAP | mPAP | Decimal | mmHg | When LABL=9, mPAP at time specified by TRLD. When LABL= 1, 2, 3 or 4 (dosing record), DV=0 mPAP=0 |
| MPAPFLD | mPAP ratio to<br>baseline (fold<br>change) | Decimal | - | When LABL=9, mPAPFLD at time specified by TRLD. When LABL= 1, 2, 3 or 4 (dosing record), DV=0 mPAPFLD=0 |
| MPAPCHG | mPAP change from baseline | Decimal | mmHg | When LABL=9, mPAPCHG at time specified by TRLD. When LABL= 1, 2, 3 or 4 (dosing record), DV=0 mPAPCHG=0 |
| EVID | Event Identification data item | Integer | - | Flag indicating whether LABL contains dosing admin info or drug concentration data. Valid values are - 1 – each dosing record for subject 0 - for all other records |

| Label | Description | Units |
|---|---|---|
| 1 | Dosing records for 0.1 mg/Kg GSK2586881 | |
| 2 | Dosing records for 0.2 mg/Kg GSK2586881 | |
| 3 | Dosing records for 0.4 mg/Kg GSK2586881 | |
| 4 | Dosing records for 0.8 mg/Kg GSK2586881 | |
| 9 | Observed hemodynamic record at time specified by TRLD; excludes NA, IS and NR, includes non-quantifiable (NQ) data | |

# 13.10. Appendix 10: Abbreviations & Trade Marks

## 13.10.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ACE2 | Angiotensin converting enzyme type 2 |
| AE | Adverse Event |
| Ang | Angiotensin |
| A&R | Analysis and Reporting |
| AUC(0-t) | Area under the concentration time curve from time zero to the time of |
| | the last quantifiable concentration |
| $AUC(0-\infty)$ | Area under the concentration time curve extrapolated to infinity |
| CI | Cardiac Index |
| CI | Confidence Interval |
| CIL | Clinical Investigative Lead |
| CL | Clearance |
| Clast | Last observed quantifiable concentration |
| Cmax | Maximum observed plasma concentration |
| CO | Cardiac Output |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CPSR | Clinical Pharmacology Study Report |
| CS | Clinical Statistics |
| CV <sub>b</sub> /CV <sub>w</sub> | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| DOB | Date of Birth |
| DP | Decimal Places |
| DQL | Data Quality Lead |
| eCRF | Electronic Case Record Form |
| GCSP | Global Clinical Safety and Pharmacovigilance |
| GSK | GlaxoSmithKline |
| IA | Interim Analysis |
| ICH | International Conference on Harmonisation |
| ICF | Informed Consent Form |
| IDSL | Integrated Data Standards Library |
| IMMS | International Modules Management System |
| IP | Investigational Product |
| IV | Intravenous |
| GUI | Guidance |
| mmHg | Millimeter of Mercury |
| mPAP | Mean Pulmonary Artery Pressure |
| NO | Nitric Oxide |
| NT-proBNP | N-terminal pro-brain natriuretic peptide |
| OSL | Operational Study Lead |
| PAH | Pulmonary Arterial Hypertension |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |

| Abbreviation | Description |
|--------------|------------------------------------------------------|
| PK | Pharmacokinetic |
| PT | Preferred Term |
| PVR | Pulmonary Vascular Resistance |
| QC | Quality Control |
| QTcF | Friderica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| RAMOS | Randomization & Medication Ordering System |
| RAS | Renin-Angiotensin-System |
| SAC | Statistical Analysis Complete |
| SAE | Serious Adverse Event |
| SD | Standard Deviation |
| SOC | System Organ Class |
| SOP | Standard Operation Procedure |
| S&P | Statistics and Programming |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |
| Tlast | Time of the last observed quantifiable concentration |
| Tmax | Time to reach Cmax |
| T1/2 | Apparent terminal half-life |
| V | Volume of distribution |

## 13.10.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies |
|---------------------------------------------------------|
| HARP |
| RANDALL NG |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| NONMEM |
| SAS |
| WinNonlin |

#### 13.11. Appendix 11: List of Data Displays

#### 13.11.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------------------------|------------|------------|
| Study Population | 1.1 to 1.n | 1.1 to 1.n |
| Efficacy | 2.1 to 2.n | 2.1 to 2.n |
| Safety | 3.1 to 3.n | 3.1 to 3.n |
| Pharmacokinetic | 4.1 to 4.n | 4.1 to 4.n |
| Population Pharmacokinetic (PopPK) | 5.1 to 5.n | 5.1 to 5.n |
| Pharmacodynamic and / or Biomarker | 6.1 to 6.n | 6.1 to 6.n |
| Pharmacokinetic / Pharmacodynamic | 7.1 to 7.n | 7.1 to 7.n |
| Section | List | ings |
| ICH Listings | 1 to x | |
| Other Listings | y to z | |

#### 13.11.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required example mock-up displays provided in Appendix 13: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------------------------|----------|----------|----------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Efficacy | EFF_Fn | EFF_Tn | EFF_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |
| Population Pharmacokinetic (PopPK) | POPPK_Fn | POPPK_Tn | POPPK_Ln |
| Pharmacodynamic and / or Biomarker | PD_Fn | PD_Tn | PD_Ln |
| Pharmacokinetic / Pharmacodynamic | PKPD_Fn | PKPD_Tn | PK/PD_Ln |

#### NOTES:

Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

#### 13.11.3. Deliverables

| Delivery | Description |
|---|---|
| DE [1] | Dose Escalation Dose 1 (Responsibility of GSK) |
| DE [2] | Dose Escalation Dose 2 (Responsibility of GSK) |
| DE [3] | Dose Escalation Dose 3 (Responsibility of GSK) |
| SAC / | Final Statistical Analysis Complete / |
| SAC(GSK) | Final Statistical Analysis Complete (Responsibility of GSK) |

## 13.11.4. Study Population Tables

| Study | Population Tab | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1.1. | Safety | ES1 | Summary of Participant Disposition for the Participant Conclusion Record | ICH E3, FDAAA, EudraCT | SAC |
| 1.2. | Screened | ES6 | Summary of Screening Status and Reasons for Screen Failure | Journal Requirements | SAC |
| 1.3. | Safety | NS1 | Summary of Number of Participants by Country and Site ID | EudraCT/Clinical Operations | SAC |
| Protoc | ol Deviation | | | | |
| 1.4. | Safety | DV1 | Summary of Important Protocol Deviations | ICH E3 | SAC |
| Popula | tion Analysed | | | | |
| 1.5. | Safety | SP1 | Summary of Study Populations | IDSL | SAC |
| Demog | raphic and Bas | eline Characteris | tics | | |
| 1.6. | Safety | DM1 | Summary of Demographic Characteristics | ICH E3, FDAAA, EudraCT | SAC |
| 1.7. | Safety | DM11 | Summary of Age Ranges | EudraCT | SAC |
| 1.8. | Safety | DM5 | Summary of Race and Racial Combinations | ICH E3, FDA, FDAAA, EudraCT | SAC |
| 1.9. | Safety | POP_T1 | Summary of Baseline Characteristics | Include Functional Class (I, II, III) (frequencies) and 6MWD (summary stats) and PAH underlying causes (frequencies) by dose group and overall | SAC |

| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| Prior a | nd Concomitan | t Medications | | | |
| 1.10. | Safety | MH1 | Summary of Past Medical Conditions | ICH E3 | SAC |
| 1.11. | Safety | MH1 | Summary of Current Medical Conditions | ICH E3 Separate summaries for Current & Past conditions, if collected. | SAC |
| 1.12. | Safety | CM1 | Summary of Concomitant Medications | ICH E3 | SAC |
| 1.13. | Safety | CM1 | Summary of Concomitant Medications for PAH | Will be based on a spreadsheet review by the medical monitor to flag those records within the conmed dataset that were applicable to PAH. This flag will be read in and merged when creating the CMANAL dataset. One review prior to DBF for pre-programming and a final review (quick turnaround) at DBF. | SAC |
| Exposu | re and Treatmen | t Compliance | | | |
| 1.14. | Safety | EX3 | Listing of Exposure to Study Treatment | ICH E3 | SAC |

# 13.11.5. Safety Tables

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events (AEs) | | | | |
| 3.1. | Safety | AE1CP | Summary of All Adverse Events by System Organ Class and Preferred Term | ICH E3 | SAC |
| 3.2. | Safety | AE1CP | Summary All Drug-Related Adverse Events by System Organ Class and Preferred Term/by Overall Frequency | ICH E3 | SAC |
| Serious | and Other Sig | nificant Adverse | Events | | |
| 3.3. | Safety | AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Participants and Occurrences) | FDAAA, EudraCT | SAC |
| ECG | | | | | |
| 3.4. | Safety | EG1 | Summary of ECG Findings | IDSL | SAC |
| 3.5. | Safety | EG2 | Summary of Change from Baseline in ECG Values by Visit | IDSL | SAC |
| 3.6. | Safety | CP_EG11 | Frequency of ECG Values by Pre-Specified PCI Categories | Categories as per PCI details in Section 13.7.2 | SAC |
| 3.7. | Safety | CP_EG12 | Frequency of Change from Baseline ECG Values by Pre-<br>Specified PCI Categories | Categories as per PCI details in Section 13.7.2 | SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Vital Sig | gns | | | | |
| 3.8. | Safety | VS1 | Summary of Change from Baseline in Vital Signs | ICH E3 | SAC |
| Pulse O | ximetry | | | | |
| 3.9. | Safety | VS1 | Summary of Oxygen Saturation | Collected at same timepoints as vital signs (but no triplicates at pre-dose) | SAC |
| Immund | Immunogenicity | | | | |
| 3.10. | Safety | IMM1 | Summary of Positive Immunogenicity Results | Results will be categorised by visit (Day 7, Day 28) and dose group within the table. | SAC |

## 13.11.6. Safety Figures

| Safety: | Safety: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events | | | | |
| 3.1. | Safety | SAF_F1 | Summary of Change from Baseline (95% CI) in Systolic Blood Pressure by Dose Group | Data from VITALS dataset. See example, x-axis will be post-dose timepoint with each dose group mean ±95% CI plotted (dose groups offset) Include a horizontal dashed grey line at zero. Please use symbols as indicated in Section 5.1 | SAC |
| 3.2. | Safety | SAF_F1 | Summary of Change from Baseline (95% CI) in Diastolic Blood Pressure by Dose Group | Data from VITALS dataset. See example, x-axis will be post-dose timepoint with each dose group mean ±95% CI plotted (dose groups offset) Include a horizontal dashed grey line at zero. Please use symbols as indicated in Section 5.1 | SAC |
| 3.3. | Safety | SAF_F1 | Summary of Change from Baseline (95% CI) in Heart Rate by Dose Group | Data from VITALS dataset. See example: x-axis will be post-dose timepoint with each dose group mean ±95% CI plotted (dose groups offset) Include a horizontal dashed grey line at zero. Please use symbols as indicated in Section 5.1 | SAC |

| Safety: | Safety: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.4. | Safety | SAF_F2 | Summary of Individual Systolic Blood Pressure by Dose Group | Data from VITALS dataset. See example: One plot per dose group, with all subject profiles on each dose group plot, 4 pages per output | SAC |
| 3.5. | Safety | SAF_F2 | Summary of Individual Diastolic Blood Pressure by Dose Group | Data from VITALS dataset. See example: One plot per dose group, with all subject profiles on each dose group plot, 4 pages per output | SAC |
| 3.6. | Safety | SAF_F2 | Summary of Individual Heart Rate by Dose Group | Data from VITALS dataset. See example: One plot per dose group, with all subject profiles on each dose group plot, 4 pages per output | SAC |
### 13.11.7. Pharmacokinetic Tables

| Pharma | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Con | centration Data | a | | | |
| 4.1. | PK | PKCT1 (PK01) | Summary of GSK2586881 Pharmacokinetic Concentration-Time Data (ng/mL) | By dose group | SAC |
| PK Para | ameter Data | | | | |
| 4.2. | PK | PKPT1 (PK03) | Summary Statistics of Derived Plasma GSK2586881<br>Pharmacokinetic Parameters | By dose group. See Section 9.1.1.2 for full list of parameters to be expected | SAC |
| 4.3. | PK | PKPT3 (PK05) | Summary Statistics of Log-Transformed Derived Plasma<br>GSK2586881 Pharmacokinetic Parameters | By dose group. See Section 9.1.1.2 for full list of parameters to be expected (Tmax, lambda_x variables, #pts and R2 not included) | SAC |

## 13.11.8. Pharmacokinetic Figures

| Pharma | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Con | centration | | | | |
| 4.1. | PK | PKCF1P<br>(PK16a) | Individual GSK2586881 Plasma Concentration–Time Plots (Linear and Semi-log) | By Subject plots | SAC |
| 4.2. | PK | PKCF6 (PK24) | Individual GSK2586881 Plasma Concentration–Time Plot (Linear and Semi-log) | Page by dose group, all subjects on a plot for each dose group | SAC |
| 4.3. | PK | PKCF2 (PK17) | Mean Plasma GSK2586881 Concentration-Time Plot (Linear and Semi-Log) | Include a legend for dose groups | SAC |
| 4.4. | PK | PKCF3 (PK18) | Median Plasma GSK2586881 Concentration-Time Plot | Include a legend for dose groups | SAC |
| 4.5. | PK | (PK28) | Plot of Individual (+Geometric Mean and 95% CIs) GSK2586881<br>Cmax versus Dose | | SAC |
| 4.6. | PK | (PK28) | Plot of Individual (+Geometric Mean and 95% CIs) GSK2586881 AUC(0-t) versus Dose | | SAC |
| 4.7. | PK | (PK28) | Plot of Individual (+Geometric Mean and 95% CIs) GSK2586881 AUC(0-inf) versus Dose | | SAC |

# 13.11.9. Pharmacodynamic and Biomarker Tables

| Pharma | Pharmacodynamic (and or Biomarker): Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Hemod | ynamics | | | | |
| 6.1. | Evaluable | PD_T1 (or<br>modify PFT1 &<br>PFT2) | Summary of Pulmonary Hemodynamics (Absolute) | Interim Tables Include PVR, CO mPAP & CI only for dose group being assessed at the time (can be indicated in the title 'Dose Group = xx mg/kg') Provide second page with geometric means etc (from log-transformation) SAC Table By dose group and endpoint (x9 PVR, CO, mPAP, Right Atrial Pressure etc). n[1] in mock not required for Hemodynamic endpoints. Log-transformed summary to be included as a second page for each parameter (see mock). Timepoints are Pre-dose, 1h, 2h and 4h. | DE[1],<br>DE[2],<br>DE[3] &<br>SAC |

| Pharma | acodynamic (aı | nd or Biomarker): | Tables | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 6.2. | Evaluable | PD_T1 (or<br>modify PFT1 &<br>PFT2) | Summary of Change from Baseline in Pulmonary Hemodynamics | Interim Tables Include PVR, CO mPAP & CI only for dose group being assessed at the time (can be indicated in the title 'Dose Group = xx mg/kg') Provide second page with geometric means etc (from log-transformation) SAC Table By dose group and endpoint (x9 PVR, CO, mPAP, Right Atrial Pressure etc). Pre-dose excluded. n[1] in mock not required for Hemodynamic endpoints. Log-transformed summary to be included as a second page for each parameter (see mock). Timepoints are 1h, 2h and 4h. | DE[1],<br>DE[2],<br>DE[3] &<br>SAC |
| 6.3. | Evaluable | PD_T3 | Summary of Statistical Analysis of PVR, CO, mPAP and CI | Interim Tables Utilising Bayesian version of repeated measures mixed effect modelling results for dose group(s) of interest at the time. Posterior probabilities to be included, see Section 7.1.5.1. SAC table As above, with consideration to all dose groups, discuss with team to ensure probabilities of interest are displayed as further probabilities may be required in addition to those quoted in Section 7.1.5.1. | DE[1],<br>DE[2],<br>DE[3],<br>SAC (GSK) |

| Pharma | Pharmacodynamic (and or Biomarker): Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| RAS | | | | | |
| 6.4. | Evaluable | PD_T1 (or<br>modify PFT1 &<br>PFT2) | Summary of Venous (Systemic) RAS<br>Peptides (Absolute Data) | By dose group and analyte. Log-transformed summary to be included as a second page for each parameter. To include <b>Angll, Ang(1-7), Ang(1-5)</b> . Timepoints are Pre-dose, 0.5h, 1h, 2h, 4h, 8h, 24h and Day(7-14) FU | SAC |
| 6.5. | Evaluable | PD_T1 (or<br>modify PFT1 &<br>PFT2) | Summary of Pulmonary Wedge RAS<br>Peptides (Absolute Data) | By dose group and analyte. Log-transformed summary to be included as a second page for each parameter. To include <b>Ang II</b> , <b>Ang(1-7)</b> , <b>Ang(1-5)</b> . Timepoints are Pre-dose, 1h, 2h and 4h only. | SAC |
| 6.6. | Evaluable | PD_T1 (or<br>modify PFT1 &<br>PFT2) | Summary of Change from Baseline in Venous (Systemic) RAS Peptides | By dose group and analyte. Log-transformed summary to be included as a second page for each parameter. To include <b>Angll</b> , <b>Ang(1-7)</b> , <b>Ang(1-5)</b> . Timepoints are 0.5h, 1h, 2h, 4h, 8h, 24h and Day(7-14) FU | SAC |
| 6.7. | Evaluable | PD_T1 (or<br>modify PFT1 &<br>PFT2) | Summary of Change from Baseline in Pulmonary Wedge RAS Peptides | By dose group and analyte. Log-transformed summary to be included as a second page for each parameter. To include <b>Ang II</b> , <b>Ang(1-7)</b> , <b>Ang(1-5)</b> . Timepoints are 1h, 2h and 4h only. | SAC |
| 6.8. | Evaluable | PD_T2 | Summary of Venous (Systemic) RAS<br>AngII/Ang(1-7) Ratio | By dose group. Log-transformed summary to be included as a second page. Timepoints are Pre-dose, 0.5h, 1h, 2h, 4h, 8h, 24h and Day(7-14) FU | SAC |
| 6.9. | Evaluable | PD_T2 | Summary of Pulmonary Wedge RAS<br>AngII/Ang(1-7) Ratio | By dose group. Log-transformed summary to be included as a second page. Timepoints are Pre-dose, 1h, 2h, 4h | SAC |

| Pharma | Pharmacodynamic (and or Biomarker): Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Other E | Biomarkers | | | | |
| 6.10. | Evaluable | PD_T1 (or<br>modify PFT1 &<br>PFT2) | Summary of Disease Activity<br>Biomarkers (Absolute Data) | By dose group and analyte. Log-transformed summary to be included as a second page for each parameter. To include NT pro-BNP, serum NO, cardiac tropinin I. Timepoints are Pre-dose, 2h, 4h and 24h only. | SAC |
| 6.11. | Evaluable | PD_T1 (or<br>modify PFT1 &<br>PFT2) | Summary of Change from Baseline in Disease Activity Biomarkers | By dose group and analyte. Log-transformed summary to be included as a second page for each parameter. To include NT pro-BNP, serum NO, cardiac tropinin I. Timepoints are 2h, 4h and 24h only. | SAC |

## 13.11.10. Pharmacodynamic and Biomarker Figures

| Pharma | Pharmacodynamic (and or Biomarker): Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Hemodynamics | | | | | |
| 6.1. | Evaluable | PD_F3a | Individual Subject Profiles of Pulmonary<br>Hemodynamics (Absolute) | Interim Plots: All subjects on one plot. Page by endpoint CO, PVR, mPAP and CI. Include 'Dose Group = XX' within title Include a second page (similar for PD_F7) that displays the dose group profiles from 206246 side by side with the data from previous ISS study – for each parameter SAC Plots All subjects on one plot. One page per dose group. Page also by endpoint CO, PVR, mPAP and CI only. Include a second page with log10 axes. | DE[1], DE[2],<br>DE[3]<br>& SAC |
| 6.2. | Evaluable | PD_F1 | Summary of Pulmonary Hemodynamics (Absolute) | X-axis will be timepoints Pre-dose, 1h, 2h, 4h. Y-axis will be mean endpoint including 95% CI, by treatment groups (add to legend). Offset doses at each timepoint. Page by endpoint CO, PVR, mPAP and CI only Present geometric means and 95% CIs on second page. Please use symbols as indicated in Section 5.1 | SAC |

| Pharma | Pharmacodynamic (and or Biomarker): Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 6.3. | Evaluable | PD_F2 | Summary of Change from Baseline in Pulmonary Hemodynamics | X-axis will be timepoints 1h, 2h, 4h. Y-axis will be mean endpoint including 95% CI, by treatment groups (add to legend). Offset doses at each timepoint. Page by endpoint CO, PVR, mPAP and CI only Present geometric means and 95% CIs on second page. Please use symbols as indicated in Section 5.1 | SAC |
| 6.4. | Evaluable | PD_F4 | Linear Regression Plots for Post-dose<br>Changes from Baseline vs Dose in PVR, CO,<br>mPAP and CI | To include data from all dose groups (similar to PD_F4 but with data points plotted for 0.8 mg/kg also). One page per timepoint (1h, 2h and 4h) | SAC |

| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| RAS Bi | omarkers | • | | | . ,, |
| 6.5. | Evaluable | PD_F3b | Individual Subject Profiles of Venous<br>(Systemic) RAS Biomarkers | Interim Plots (as required based on data availability) All subjects on one plot, one page per dose group and endpoint. Include a second page (similar to PD_F8) that displays the dose group profiles from 206246 side by side with the data from previous ISS study – primarily for AnglI and Ang(1-7). SAC Plot All subjects on one plot, one page per dose group. AnglI x 4 pages, Ang(1-5) x 4 pages, Ang(1-7) x 4 pages. Timepoints are Pre-dose, 0.5h, 1h, 2h, 4h, 8h, 24h and Day(7-14) FU Include a second page with log10 axes for each endpoint/dose group | <b>DE[1], DE[2</b><br><b>DE[3]</b><br>& SAC |
| 6.6. | Evaluable | PD_F3b | Individual Subject profiles of Pulmonary<br>Wedge RAS Biomarkers | All subjects on one plot, one page per dose group: Ang II x 4 pages, Ang(1-5) x 4 pages, Ang(1-7) x 4 pages, Ang II/Ang(1-7) x 4 pages. Timepoints are Pre-dose, 1h, 2h and 4h only. Include a second page with log10 axes for each endpoint/dose group. | SAC |

| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 6.7. | Evaluable | PD_F1 | Summary of Venous (Systemic) RAS<br>Biomarkers (Absolute) | X-axis will be timepoints Pre-dose, 0.08h, 0.5h, 1h, 2h, 4h, 8h, 24h, FU7-14. Y-axis will be <b>geometric</b> mean RAS including 95% CI, by dose groups (add to legend). One page per endpoint (4 x RAS endpoints). Presenting geometric means from log-transformed data (see matching table). Include Angll, Ang(1-7), Ang(1-5) and Angll/Ang(1-7) Please use symbols as indicated in Section 5.1 | SAC |
| 6.8. | Evaluable | PD_F1 | Summary of Pulmonary Wedge RAS<br>Biomarkers (Absolute) | X-axis will be timepoints Pre-dose, 1h, 2h, 4h. Y-axis will be <b>geometric</b> RAS including 95% CI, by dose groups (add to legend). One page per endpoint (4 x RAS endpoints). Presenting geometric means from log-transformed data (see matching table). Include Angll, Ang(1-7), Ang(1-5) and Angll/Ang(1-7) Please use symbols as indicated in Section 5.1 | SAC |
| 6.9. | Evaluable | PD_F5 | Correlation plot for Venous (Systemic) RAS Biomarkers | Scatter plot of Ang II vs Ang(1-7) on page 1, Ang II vs Ang(1-5) on page 2 and Ang(1-5) vs Ang(1-7) on page 3. Venous RAS timepoints. To be plotted on log-log scales. Please provide clear dose/timepoint labels within the legend, mock-up is basic example only. | SAC |

| Pharma | acodynamic (ar | nd or Biomarker): | Figures | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 6.10. | Evaluable | PD_F5 | Correlation plot for Pulmonary Wedge RAS<br>Biomarkers | Scatter plot of Ang II vs Ang(1-7) on page 1, Ang II vs Ang(1-5) on page 2 and Ang(1-5) vs Ang(1-7) on page 3. Pulmonary wedge RAS timepoints. To be plotted on log-log scales. Please provide clear dose/timepoint labels within the legend, mock-up is basic example only. | SAC |
| Diseas | e Activity Biom | arkers | | | |
| 6.11. | Evaluable | PD_F1 | Summary of Disease Activity Biomarkers (Absolute) | X-axis will be timepoints Pre-dose, 2h, 4h, 24h. Y-axis will be <b>geometric</b> mean endpoint including 95% CI, by treatment groups (add to legend). One page per endpoint (3 x endpoints) Presenting geometric means from log-transformed data (see matching table). Please use symbols as indicated in Section 5.1 | SAC |
| 6.12. | Evaluable | PD_F3b | Individual Subject profiles of Disease Activity<br>Biomarkers | All subjects on one plot, one page per dose group: NT pro-BNP x 4, NO x 4 and cardiac troponin I x 4 pages. Include a second page with log10 axes for each endpoint/dose group. | SAC |
| RAS Bi | omarkers vs H | emodynamics | | , | |
| 6.13. | Evaluable | PD_F6 | Scatter Plot (log-log) of Venous (Systemic)<br>RAS Peptides (Ang II, Ang(1-5) and Ang(1-7))<br>vs PVR | 3 pages, 1 for each RAS, 4 dose groups on each page, dose/timepoint indicated in legend. Timepoints of interest based on PVR. Log-log axes Please provide clear dose/timepoint labels within the legend, mock-up is basic example only. | SAC |

| Pharmacodynamic (and or Biomarker): Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 6.14. | Evaluable | PD_F6 | Scatter Plot (log-log) of Venous (Systemic)<br>RAS Peptides (Ang II, Ang(1-5) and Ang(1-7))<br>vs CO | 3 pages, 1 for each RAS, 4 dose groups on each page, dose/timepoint indicated in legend. Timepoints of interest based on CO. Log-log axes Please provide clear dose/timepoint labels within the legend, mock-up is basic example only. | SAC |
| 6.15. | Evaluable | PD_F6 | Scatter Plot (Semi-log) of Venous (Systemic)<br>RAS Peptides (Ang II, Ang(1-5) and Ang(1-7))<br>vs mPAP | 3 pages, 1 for each RAS, 4 dose groups on each page, dose/timepoint indicated in legend. Timepoints of interest based on mPAP. Log-log axes Please provide clear dose/timepoint labels within the legend, mock-up is basic example only. | SAC |
| 6.16. | Evaluable | PD_F6 | Scatter Plot (log-log) of Venous (Systemic)<br>RAS Peptides (Ang II, Ang(1-5) and Ang(1-7))<br>vs CI | 3 pages, 1 for each RAS, 4 dose groups on each page, dose/timepoint indicated in legend. Timepoints of interest based on CI. Log-log axes Please provide clear dose/timepoint labels within the legend, mock-up is basic example only. | SAC |
| 6.17. | Evaluable | PD_F6 | Scatter Plot (Semi-log) of Pulmonary Wedge<br>RAS Peptides (Ang II, Ang(1-5) and Ang(1-7))<br>vs PVR | 3 pages, 1 for each RAS, 4 dose groups on each page, dose/timepoint indicated in legend. Timepoints of interest based on PVR. Log-log axes Please provide clear dose/timepoint labels within the legend, mock-up is basic example only. | SAC |

| Pharma | Pharmacodynamic (and or Biomarker): Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 6.18. | Evaluable | PD_F6 | Scatter Plot (Semi-log) of Pulmonary Wedge<br>RAS Peptides (Ang II, Ang(1-5) and Ang(1-7))<br>vs CO | 3 pages, 1 for each RAS, 4 dose groups on each page, dose/timepoint indicated in legend. Timepoints of interest based on CO. Log-log axes Please provide clear dose/timepoint labels within the legend, mock-up is basic example only. | SAC |
| 6.19. | Evaluable | PD_F6 | Scatter Plot (Semi-log) of Pulmonary Wedge<br>RAS Peptides (Ang II, Ang(1-5) and Ang(1-7))<br>vs mPAP | 3 pages, 1 for each RAS, 4 dose groups on each page, dose/timepoint indicated in legend. Timepoints of interest based on mPAP. Log-log axes Please provide clear dose/timepoint labels within the legend, mock-up is basic example only. | SAC |
| 6.20. | Evaluable | PD_F6 | Scatter Plot (Semi-log) of Pulmonary Wedge<br>RAS Peptides (Ang II, Ang(1-5) and Ang(1-7))<br>vs CI | 3 pages, 1 for each RAS, 4 dose groups on each page, dose/timepoint indicated in legend. Timepoints of interest based on CI. Log-log axes Please provide clear dose/timepoint labels within the legend, mock-up is basic example only. | SAC |

## 13.11.11. Pharmacokinetic / Pharmacodynamic and Biomarker Figures

| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| PK / RAS Peptides | | | | | |
| 7.1. | PK | PK_F1 | Scatter plot (Log-log) of PK Concentration vs<br>Venous (Systemic) Ang II, Ang(1-5), Ang(1-7)<br>and AngII/Ang(1-7) | Scatter plot of PK conc vs Ang II on page 1, PK conc vs Ang(1-5) on page 2, PK conc vs Ang(1-7) on page 3 and PK conc vs AngII/Ang(1-7) on page 4. Timepoints of interest based on PK. To be plotted on log-log scales. Please provide clear dose/timepoint labels within the legend, mock-up is basic example only. Note: For PK/PD plots only, PK concentration data recorded as NQ can be imputed following the same method for biomarker data i.e., replace with ½ LLQ. The imputed variable for PK should be available in the PKCNC dataset. See Section 13.4.3 Footnote to include: 'Note: Values below Lower Limit of Quantification (LLQ) replaced with ½ LLQ. LLQ for PK concentration = xx ng/mL, LLQ for AngII = xx pg/mL, LLQ for Ang(1-5) = xx pg/mL and LLQ for Ang(1-7) = xx pg/mL.' | SAC |

| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 7.2. | PK | PK_F1 | Scatter plot (Log-log) of PK Concentration vs<br>Pulmonary Wedge Ang II, Ang(1-5), Ang(1-7)<br>and AngII/Ang(1-7) | Scatter plot of PK conc vs Ang II on page 1, PK conc vs Ang(1-5) on page 2, PK conc vs Ang(1-7) on page 3 and PK conc vs AngII/Ang(1-7) on page 4. Timepoints of interest based on Pulmonary Wedge RAS. To be plotted on log-log scales. Please provide clear dose/timepoint labels within the legend, mock-up is basic example only. Note: For PK/PD plots only, PK concentration data recorded as NQ can be imputed following the same method for biomarker data i.e., replace with ½ LLQ. The imputed variable for PK should be available in the PKCNC dataset. See Section 13.4.3 Footnote to include: 'Note: Values below Lower Limit of Quantification (LLQ) replaced with ½ LLQ. LLQ for PK concentration = xx ng/mL, LLQ for AngII = xx pg/mL, LLQ for Ang(1-5) = xx pg/mL and LLQ for Ang(1-7) = xx pg/mL.' | SAC |

| Pharmacokinetic / Pharmacodynamic: Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 7.3. | PK | PK_F1 | Scatter Plot (Log-log) of PK Concentration vs<br>PVR, CO, mPAP and CI | Scatter plot of PK conc vs PVR on page 1, PK conc vs CO on page 2, PK conc vs mPAP on page 3 and PK conc vs CI on page 4. Timepoints of interest based on hemodynamics. To be plotted on log-log scales. Please provide clear dose/timepoint labels within the legend, mock-up is basic example only. Note: For PK/PD plots only, PK concentration data recorded as NQ can be imputed following the same method for biomarker data i.e., replace with ½ LLQ. The imputed variable for PK should be available in the PKCNC dataset. See Section 13.4.3. Footnote to include: 'Note: Values below Lower Limit of Quantification (LLQ) replaced with ½ LLQ. LLQ for PK concentration = xx ng/mL.' | SAC |

## 13.11.12. ICH Listings

| ICH: Li | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1. | Screened | ES7 | Listing of Reasons for Screen Failure | Journal Guidelines | SAC |
| 2. | Safety | ES2 | Listing of Reasons for Study Withdrawal | ICH E3 | SAC |
| 3. | Safety | TA1 | Listing of Planned and Actual Treatments | IDSL | SAC |
| Protoc | ol Deviations | | | | |
| 4. | Safety | DV2 | Listing of Important Protocol Deviations | ICH E3 | SAC |
| 5. | Safety | IE3 | Listing of Participants with Inclusion/Exclusion Criteria Deviations | ICH E3 | SAC |
| Popula | tions Analysed | | | | |
| 6. | Safety | SP3 | Listing of Participants Excluded from Any Population | ICH E3 | SAC |
| Demog | raphic and Bas | eline Characteris | tics | | |
| 7. | Safety | DM2 | Listing of Demographic Characteristics | ICH E3 | SAC |
| 8. | Safety | DM9 | Listing of Race | ICH E3 | SAC |
| Prior a | nd Concomitan | t Medications | | | |
| 9. | Safety | CP_CM3 | Listing of Concomitant Medications | IDSL | SAC |
| Exposi | ure and Treatme | ent Compliance | | | |
| 10. | Safety | EX3 | Listing of Exposure Data | ICH E3 | SAC |
| Advers | e Events | | | | |
| 11. | Safety | AE8CP | Listing of All Adverse Events | ICH E3 | SAC |
| 12. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events | ICH E3 | SAC |

| ICH: Li | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Serious | s and Other Sig | nificant Adverse | Events | | |
| 13. | Safety | AE8CPa | Listing of Serious Adverse Events | ICH E3 | SAC |
| 14. | Safety | AECP8 | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment | ICH E3 | SAC |
| All Lab | oratory | | | | |
| 15. | Safety | LB5 | Listing of All Laboratory Data for Participants with Any Value of Potential Clinical Importance/Outside Normal Range | ICH E3 | SAC |
| 16. | Safety | LB5 | Listing of Laboratory Values of Potential Clinical Importance | | SAC |
| ECG | | | | | |
| 17. | Safety | EG3/CP_EG3 | Listing of All ECG Values for Participants with Any Value of Potential Clinical Importance | IDSL | SAC |
| 18. | Safety | EG3/CP_EG3 | Listing of ECG Values of Potential Clinical Importance | IDSL | SAC |
| 19. | Safety | EG5/CP_EG5 | Listing of All ECG Findings for Participants with an Abnormal ECG Finding | IDSL | SAC |
| 20. | Safety | EG5/CP_EG5 | Listing of Abnormal ECG Findings | IDSL | SAC |
| Vital Si | gns | | | | |
| 21. | Safety | VS4 | Listing of All Vital Signs Data for Participants with Any Value of Potential Clinical Importance | IDSL | SAC |
| 22. | Safety | VS4 | Listing of Vital Signs of Potential Clinical Importance | IDSL | SAC |

## 13.11.13. Non-ICH Listings

| Non-IC | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Baselin | e Characterist | ics | | | |
| 23. | Safety | POP_L1 | Listing of Baseline Characteristics | | SAC |
| Pharma | acodynamic | | | | |
| 24. | Safety | PD_L2 | Listing of Hemodynamic Endpoints | Interim Listings: Produce for relevant dose group. Include % change from baseline (presented as a ratio to baseline based on back-transformed data) SAC Listing: Produce for all dose groups. Include % change from baseline (presented as a ratio to baseline based on back-transformed data) | DE[1],<br>DE[2].<br>DE[3]<br>& SAC |
| 25. | Safety | PFT8 | Listing of Oxygen Saturation | Follow PFT8 IDSL format, replacing last 4 columns with Oxygen Saturation endpoint. | SAC |
| Biomar | kers | | | | |
| 26. | Safety | PD_L1 | Listing of Venous (Systemic) RAS Peptides | See non-standard example PD_L1. To include AngII, Ang(1-5) and Ang(1-7) | SAC |
| 27. | Safety | PD_L1 | Listing of Pulmonary Wedge RAS Peptides | See non-standard example PD_L1 (4 timepoints only) To include AngII, Ang(1-5) and Ang(1-7) | SAC |
| 28. | Safety | PD_L1 | Listing of Disease Biomarkers | See non-standard example PD_L1 (4 timepoints only) | SAC |
| Immun | ogenicity | | ' | | • |
| 29. | Safety | IMM2 | Listing of Immunogenicity | | SAC |

| Non-ICI | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | |
| PK | | | | | |
| 30. | PK | PKCL1P<br>(PK07) | Listing of GSK2586881 Plasma<br>Pharmacokinetic Concentration—<br>Time Data | | SAC |
| 31. | PK | PKPL1P<br>(PK13) | Listing of Derived GSK2586881 Plasma Pharmacokinetic Parameters | See Section 9.1.1.2 for list of parameters. To include lambda_z and the additionally the first point, last point and number of points used in the determination of lambda_z for listings and R squared. | SAC |

## 13.12. Appendix 13: Example Mock Shells for Data Displays

Data Display Specification will be made available on Request